CLINICAL TRIAL: NCT01209078
Title: A Randomized, Double Blind, Double Dummy Multicenter Phase IIa Study to Assess Safety, Tolerability and Efficacy of GSK1322322 Versus Linezolid in the Treatment of Acute Bacterial Skin and Skin Structure Infection
Brief Title: GSK1322322 Versus Linezolid in the Treatment of Acute Bacterial Skin and Skin Structure Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113414
Record Dates: First submitted 2010-09-14; First posted 2010-09-24 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-09

CONDITIONS: Skin Infections, Bacterial
Keywords: methicillin-resistant Staphylococcus aureus; linezolid; repeat dose; GSK1322322
MeSH Terms: conditions — Cellulitis | interventions — GSK1322322; Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regimen 1 (Experimental): GSK1322322 1500mg and Placebo Linezolid given twice a day (BID) for 10 days
  Interventions: Drug: GSK1322322; Drug: Linezolid placebo
- Regimen 2 (Active Comparator): Linezolid 600mg and placebo GSK1322322 given BID for 10 days
  Interventions: Drug: Linezolid; Drug: GSK1322322 placebo

INTERVENTIONS:
Drug: GSK1322322 — GSK1322322 1500mg BID
  Arms: Regimen 1
Drug: Linezolid — Linezolid 600mg
  Arms: Regimen 2
Drug: GSK1322322 placebo — Placebo
  Arms: Regimen 2
Drug: Linezolid placebo — placebo
  Arms: Regimen 1

SUMMARY:
This study will determine the safety, tolerability and efficacy of GSK1322322 verses Linezolid in subjects with Acute Bacterial Skin and Skin Structure Infection (ABSSSI).

DETAILED DESCRIPTION:
This is a phase IIa, multicenter, randomized, parallel group, double-blind, double dummy study to assess the safety, tolerability, and efficacy of GSK1322322 when given as 1500mg twice daily over a 10-day period versus linezolid (600mg twice daily for 10 days) in adults with suspected Gram positive Acute Bacterial Skin and Skin Structure Infection who are not currently receiving antibacterial therapy. Subjects will be randomized (2:1) to GSK1322322 or linezolid. This study consists of a screening visit, a 10-day treatment period, and follow-up evaluations 7 and 28 days following the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject age 18 years or older at the time of signing the informed consent
* Male subjects must agree to use one of the contraception methods listed
* A female is eligible to enter and participate in this study if she is of non-childbearing potential
* The subject has a diagnosis of ABSSSI defined as one of the following: wound infection with cellulitis that has developed within 30 days of surgery or trauma; abscess with cellulitis, or cellulitis that has developed in no more than 7 days before enrollment with worsening over the past 48 hours OR in the investigator's opinion the patient's condition warrants systemic oral antibiotic therapy
* The subject has at least 2 additional signs and symptoms of skin infection: purulence, erythema with or without induration, fluctuation, heat/localized warmth, and pain/tenderness
* The subject has at least 1 systemic marker of infection: Lymphadenopathy, Fever (>38 degrees Celsius), White Blood Cell elevation, or Creatinine Reactive Protein (CRP) >Upper Limit of Normal (ULN)
* The subject has given written, informed, dated consent to participate in the study
* QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) < 2xULN; and bilirubin < 1.0xULN

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* The subject has been diagnosed with Acquired immune deficiency syndrome (AIDS)
* Body mass index (BMI) >40 kg/m2
* The subject has demonstrated a previous hypersensitivity reaction to GSK1322322, or to oxazolidinones
* The subject has a secondarily infected animal/human bite
* The subject has a chronic ulcerative lesion that is likely to be polymicrobial or caused by anaerobic organisms and unlikely to have Staphylococcus aureus or Streptococcus pyogenes as the causative agent
* The subject has an underlying skin disease, such as pre-existing eczematous dermatitis, with clinical evidence of secondary infection
* The subject has an infection that would normally have a high cure rate after surgical incision alone
* The subject has a bacterial skin infection which, due to the extent, depth or severity of clinical presentation, in the opinion of the investigator, cannot be appropriately treated by an oral antibiotic
* The subject has received more than one dose of treatment with a systemic and/or topical antibacterial within 7 days
* The subject is currently receiving vasopressors
* The subject is currently receiving adrenergic agents
* The subject is currently receiving serotonergic reuptake inhibitors
* The subject is currently receiving monoamine oxidase inhibitors
* The subject has a documented clinical history of pseudomembranous colitis
* The subject has known, pre-existing myelosuppression, or a history of myelosuppression with prior linezolid use, or is currently receiving a medication that produces bone marrow suppression
* The subject has a history of seizures
* The subject has a history of severe renal failure and is undergoing dialysis
* The subject has a serious underlying disease that could be imminently life-threatening
* The subject has been previously enrolled in this study
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product
* Subject is unable to discontinue the use of prescription drugs listed in the protocol or non-prescription drugs, including vitamins, herbal and dietary supplements prior to the first dose of study medication through the first follow up visit
* Lactating females or pregnant females as determined by positive urine pregnancy test at screening or prior to dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-08-17 (Actual); Primary Completion 2011-01-18 (Actual); Study Completion 2011-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (7):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Oceanside, California
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, West Reading, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Corey R, Naderer OJ, O'Riordan WD, Dumont E, Jones LS, Kurtinecz M, Zhu JZ. Safety, tolerability, and efficacy of GSK1322322 in the treatment of acute bacterial skin and skin structure infections. Antimicrob Agents Chemother. 2014 Nov;58(11):6518-27. doi: 10.1128/AAC.03360-14. Epub 2014 Aug 18. PMID 25136015
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 113414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned on 75 male and female participants with Gram-positive acute bacterial skin and skin structure infection (ABSSSI) who were not receiving any antibacterial therapy, aged 18 years or older at eight study centers in the United States from 13 September 2010 to 20 December 2010.
Pre-assignment Details: A total of 84 participants were enrolled in the study; of which, 57 participants were randomized in a ratio of 2:1 to receive GSK1322322 1500 milligram (mg) twice a day (BID) and 27 were randomized to receive linezolid 600 mg BID for 10 days.
Groups:
- GSK1322322 1500 mg BID: Participants received oral dose of GSK1322322 1500 mg as 3 tablets of 500 mg each, BID in the morning and evening for 10 days. Blinding was maintained by administration of matching placebo capsules to linezoid in the morning and evening. The study medication was taken with 240 milliliter (mL) of water or liquid.
- Linezolid 600 mg BID: Participants received oral dose of linezolid 600 mg tablet BID in the morning and evening for 10 days. Blinding was maintained by administration of matching placebo tablets to GSK1322322 in the morning and evening. The study medication was taken with 240 mL of water or liquid.
Period: Overall Study
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Started | 57 | 27
Completed | 41 | 24
Not Completed | 16 | 3
Not completed — Adverse Event | 5 | 0
Not completed — Lost to Follow-up | 4 | 0
Not completed — Physician Decision | 5 | 2
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- GSK1322322 1500 mg BID: Participants received oral dose of GSK1322322 1500 mg as 3 tablets of 500 mg each, BID in the morning and evening for 10 days. Blinding was maintained by administration of matching placebo capsules to linezoid in the morning and evening. The study medication was taken with 240 mL of water or liquid.
- Total: Total of all reporting groups
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID | Total
Number analyzed (Participants) | 57 | 27 | 84
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.4 (11.87) | 41.5 (11.00) | 43.5 (11.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 4 | 18
  Male | 43 | 23 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 4 | 2 | 6
  White | 47 | 23 | 70
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, associated with liver injury and impaired liver function defined as alanine aminotransferase (ALT) >=3 x upper limit of normal (ULN), and total bilirubin >=2 x ULN or international normalised ratio >1.5.
Time Frame: Up to Follow-up (28 Day Follow-up, Day 40)
Population: Safety Population was defined as all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Participants
  Any AE | 49 | 20
  Any SAE | 1 | 1

2. Primary Outcome: Mean Clinical Chemistry Parameters of Albumin and Total Protein at Indicated Time Points
Description: Blood samples were obtained for analysis of albumin and total protein at Day 1, Day 4, Day 8, Day 11, 7 Day Follow-up and 28 Day Follow-up. Baseline value was defined as the assessment done on Day 1.
Time Frame: Up to Follow-up (28 Day Follow-up, Day 40)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Gram/Liter
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Gram/Liter
  Albumin, Day 1: number analyzed (Participants) | 55 | 27
  Albumin, Day 1 | 39.9 (3.41) | 40.3 (3.47)
  Albumin, Day 4: number analyzed (Participants) | 45 | 25
  Albumin, Day 4 | 40.0 (3.70) | 40.5 (2.66)
  Albumin, Day 8: number analyzed (Participants) | 44 | 24
  Albumin, Day 8 | 40.3 (4.04) | 40.4 (3.35)
  Albumin, Day 11: number analyzed (Participants) | 40 | 23
  Albumin, Day 11 | 40.9 (3.59) | 42.2 (2.83)
  Albumin, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  Albumin, 7 Day Follow-up | 41.4 (4.03) | 42.8 (3.02)
  Albumin, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  Albumin, 28 Day Follow-up | 41.5 (4.03) | 41.1 (3.04)
  Total protein, Day 1: number analyzed (Participants) | 55 | 27
  Total protein, Day 1 | 72.6 (5.86) | 72.2 (6.86)
  Total protein, Day 4: number analyzed (Participants) | 45 | 25
  Total protein, Day 4 | 72.0 (5.98) | 72.4 (6.80)
  Total protein, Day 8: number analyzed (Participants) | 44 | 24
  Total protein, Day 8 | 72.8 (5.94) | 71.3 (4.46)
  Total protein, Day 11: number analyzed (Participants) | 40 | 23
  Total protein, Day 11 | 73.2 (6.19) | 73.4 (4.58)
  Total protein, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  Total protein, 7 Day Follow-up | 73.5 (5.79) | 74.3 (6.44)
  Total protein, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  Total protein, 28 Day Follow-up | 73.2 (6.35) | 72.6 (4.42)

3. Primary Outcome: Mean Clinical Chemistry Parameters of ALT, Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Follicle Stimulating Hormone (FSH), Gamma Glutamyl Transferase (GGT), Lactate Dehydrogenase (LDH) and Creatine Kinase at Indicated Time Points
Description: Blood samples were obtained for analysis of ALT, ALP, AST, FSH, GGT, LDH and creatine kinase at Day 1, Day 4, Day 8, Day 11, 7 Day Follow-up and 28 Day Follow-up. Baseline value was defined as the assessment done on Day 1.
Time Frame: Up to Follow-up (28 Day Follow-up, Day 40)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units (IU)/Liter
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
International units (IU)/Liter
  ALP, Day 1: number analyzed (Participants) | 55 | 27
  ALP, Day 1 | 102.5 (39.65) | 97.7 (34.73)
  ALP, Day 4: number analyzed (Participants) | 45 | 25
  ALP, Day 4 | 95.0 (21.99) | 92.4 (26.32)
  ALP, Day 8: number analyzed (Participants) | 44 | 24
  ALP, Day 8 | 94.8 (21.26) | 88.2 (21.63)
  ALP, Day 11: number analyzed (Participants) | 40 | 23
  ALP, Day 11 | 95.4 (23.88) | 89.3 (19.06)
  ALP, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  ALP, 7 Day Follow-up | 95.6 (27.45) | 90.9 (22.18)
  ALP, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  ALP, 28 Day Follow-up | 95.2 (27.79) | 92.9 (29.85)
  ALT, Day 1: number analyzed (Participants) | 55 | 27
  ALT, Day 1 | 26.5 (18.55) | 27.3 (17.94)
  ALT, Day 4: number analyzed (Participants) | 45 | 25
  ALT, Day 4 | 30.1 (29.46) | 25.4 (12.11)
  ALT, Day 8: number analyzed (Participants) | 44 | 24
  ALT, Day 8 | 34.3 (30.90) | 34.0 (35.20)
  ALT, Day 11: number analyzed (Participants) | 40 | 23
  ALT, Day 11 | 39.4 (51.29) | 32.2 (30.22)
  ALT, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  ALT, 7 Day Follow-up | 37.5 (35.13) | 32.6 (25.03)
  ALT, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  ALT, 28 Day Follow-up | 28.4 (19.03) | 22.7 (10.66)
  AST, Day 1: number analyzed (Participants) | 54 | 27
  AST, Day 1 | 25.9 (14.49) | 26.3 (14.66)
  AST, Day 4: number analyzed (Participants) | 44 | 24
  AST, Day 4 | 27.3 (15.01) | 24.7 (7.69)
  AST, Day 8: number analyzed (Participants) | 44 | 24
  AST, Day 8 | 32.0 (25.19) | 29.3 (18.97)
  AST, Day 11: number analyzed (Participants) | 40 | 23
  AST, Day 11 | 34.6 (30.89) | 28.5 (15.97)
  AST, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  AST, 7 Day Follow-up | 35.5 (25.72) | 28.7 (11.37)
  AST, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  AST, 28 Day Follow-up | 30.2 (21.83) | 24.0 (10.11)
  Creatine kinase, Day 1: number analyzed (Participants) | 55 | 27
  Creatine kinase, Day 1 | 118.1 (187.13) | 191.1 (396.31)
  Creatine kinase, Day 4: number analyzed (Participants) | 45 | 25
  Creatine kinase, Day 4 | 135.2 (98.96) | 166.7 (209.06)
  Creatine kinase, Day 8: number analyzed (Participants) | 44 | 24
  Creatine kinase, Day 8 | 117.3 (71.14) | 120.3 (69.81)
  Creatine kinase, Day 11: number analyzed (Participants) | 40 | 23
  Creatine kinase, Day 11 | 135.8 (113.14) | 169.3 (200.90)
  Creatine kinase, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  Creatine kinase, 7 Day Follow-up | 204.7 (561.92) | 189.1 (235.47)
  Creatine kinase, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  Creatine kinase, 28 Day Follow-up | 155.3 (168.84) | 117.5 (64.86)
  FSH, Day 1: number analyzed (Participants) | 10 | 4
  FSH, Day 1 | 21.47 (14.585) | 16.05 (24.955)
  GGT, Day 1: number analyzed (Participants) | 55 | 27
  GGT, Day 1 | 52.9 (51.70) | 52.6 (52.17)
  GGT, Day 4: number analyzed (Participants) | 45 | 25
  GGT, Day 4 | 55.3 (56.17) | 53.4 (43.15)
  GGT, Day 8: number analyzed (Participants) | 44 | 24
  GGT, Day 8 | 57.7 (52.08) | 57.7 (45.20)
  GGT, Day 11: number analyzed (Participants) | 40 | 23
  GGT, Day 11 | 55.7 (57.22) | 53.5 (40.95)
  GGT, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  GGT, 7 Day Follow-up | 65.1 (70.73) | 52.8 (39.12)
  GGT, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  GGT, 28 Day Follow-up | 50.1 (57.09) | 42.1 (42.1)
  LDH, Day 1: number analyzed (Participants) | 1 | 0
  LDH, Day 1 | 172.0 (NA) — Only one participant was analyzed. |

4. Primary Outcome: Mean Clinical Chemistry Parameters of Creatinine, Uric Acid, Direct Bilirubin and Total Bilirubin at Indicated Time Points
Description: Blood samples were obtained for analysis of creatinine, uric acid, direct bilirubin and total bilirubin at Day 1, Day 4, Day 8, Day 11, 7 Day Follow-up and 28 Day Follow-up. Baseline value was defined as the assessment done on Day 1.
Time Frame: Up to Follow-up (28 Day Follow-up, Day 40)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles (µmol)/liter
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Micromoles (µmol)/liter
  Creatinine, Day 1: number analyzed (Participants) | 55 | 27
  Creatinine, Day 1 | 68.73 (18.911) | 66.99 (13.567)
  Creatinine, Day 4: number analyzed (Participants) | 45 | 25
  Creatinine, Day 4 | 71.48 (14.307) | 72.35 (13.123)
  Creatinine, Day 8: number analyzed (Participants) | 44 | 24
  Creatinine, Day 8 | 74.85 (16.204) | 73.42 (13.159)
  Creatinine, Day 11: number analyzed (Participants) | 40 | 23
  Creatinine, Day 11 | 74.19 (16.223) | 72.07 (12.370)
  Creatinine, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  Creatinine, 7 Day Follow-up | 70.84 (15.601) | 75.06 (21.598)
  Creatinine, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  Creatinine, 28 Day Follow-up | 72.77 (20.980) | 72.49 (13.537)
  Uric acid, Day 1: number analyzed (Participants) | 55 | 27
  Uric acid, Day 1 | 322.5 (88.53) | 293.3 (84.03)
  Uric acid, Day 4: number analyzed (Participants) | 45 | 25
  Uric acid, Day 4 | 282.2 (78.77) | 346.4 (74.21)
  Uric acid, Day 8: number analyzed (Participants) | 44 | 24
  Uric acid, Day 8 | 323.2 (73.92) | 360.4 (71.96)
  Uric acid, Day 11: number analyzed (Participants) | 40 | 23
  Uric acid, Day 11 | 370.5 (88.00) | 367.4 (84.86)
  Uric acid, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  Uric acid, 7 Day Follow-up | 386.0 (105.60) | 363.8 (97.17)
  Uric acid, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  Uric acid, 28 Day Follow-up | 358.3 (89.30) | 332.6 (79.96)
  Direct bilirubin, Day 1: number analyzed (Participants) | 55 | 27
  Direct bilirubin, Day 1 | 2.3 (1.36) | 2.5 (1.05)
  Direct bilirubin, Day 4: number analyzed (Participants) | 45 | 25
  Direct bilirubin, Day 4 | 2.4 (1.39) | 2.0 (1.00)
  Direct bilirubin, Day 8: number analyzed (Participants) | 44 | 24
  Direct bilirubin, Day 8 | 2.4 (1.24) | 1.9 (0.93)
  Direct bilirubin, Day 11: number analyzed (Participants) | 40 | 23
  Direct bilirubin, Day 11 | 2.5 (1.32) | 2.1 (0.95)
  Direct bilirubin, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  Direct bilirubin, 7 Day Follow-up | 2.6 (2.16) | 3.0 (1.18)
  Direct bilirubin, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  Direct bilirubin, 28 Day Follow-up | 2.3 (1.16) | 2.3 (0.92)
  Total bilirubin, Day 1: number analyzed (Participants) | 55 | 27
  Total bilirubin, Day 1 | 8.7 (3.87) | 8.4 (4.31)
  Total bilirubin, Day 4: number analyzed (Participants) | 45 | 25
  Total bilirubin, Day 4 | 7.3 (2.66) | 6.6 (1.87)
  Total bilirubin, Day 8: number analyzed (Participants) | 44 | 24
  Total bilirubin, Day 8 | 7.6 (3.15) | 6.6 (1.91)
  Total bilirubin, Day 11: number analyzed (Participants) | 40 | 23
  Total bilirubin, Day 11 | 8.1 (3.07) | 7.6 (2.17)
  Total bilirubin, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  Total bilirubin, 7 Day Follow-up | 8.1 (4.13) | 8.9 (4.04)
  Total bilirubin, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  Total bilirubin, 28 Day Follow-up | 8.5 (3.81) | 7.6 (3.01)

5. Primary Outcome: Mean Clinical Chemistry Parameters of Glucose, Sodium, Calcium, Potassium, Chloride, Carbon Dioxide (CO2) Content /Bicarbonate and Urea/ Blood Urea Nitrogen (BUN) at Indicated Time Points
Description: Blood samples were obtained for analysis of glucose, sodium, calcium, potassium, chloride, CO2 content /bicarbonate and urea/BUN at Day 1, Day 4, Day 8, Day 11, 7 Day Follow-up and 28 Day Follow-up. Baseline value was defined as the assessment done on Day 1.
Time Frame: Up to Follow-up (28 Day Follow-up, Day 40)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimole (mmol)/Liter
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Millimole (mmol)/Liter
  Glucose, Day 1: number analyzed (Participants) | 55 | 27
  Glucose, Day 1 | 6.21 (2.385) | 6.63 (5.652)
  Glucose, Day 4: number analyzed (Participants) | 45 | 25
  Glucose, Day 4 | 6.13 (2.459) | 6.77 (5.834)
  Glucose, Day 8: number analyzed (Participants) | 44 | 24
  Glucose, Day 8 | 5.94 (1.473) | 5.77 (1.618)
  Glucose, Day 11: number analyzed (Participants) | 40 | 23
  Glucose, Day 11 | 6.27 (2.025) | 6.65 (3.355)
  Glucose, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  Glucose, 7 Day Follow-up | 5.96 (1.607) | 6.40 (2.212)
  Glucose, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  Glucose, 28 Day Follow-up | 6.10 (1.487) | 6.76 (3.068)
  Sodium, Day 1: number analyzed (Participants) | 55 | 27
  Sodium, Day 1 | 138.3 (2.49) | 138.3 (3.17)
  Sodium, Day 4: number analyzed (Participants) | 45 | 25
  Sodium, Day 4 | 137.3 (3.07) | 138.3 (1.96)
  Sodium, Day 8: number analyzed (Participants) | 44 | 24
  Sodium, Day 8 | 137.8 (1.99) | 138.4 (3.11)
  Sodium, Day 11: number analyzed (Participants) | 40 | 23
  Sodium, Day 11 | 138.6 (2.11) | 138.2 (2.79)
  Sodium, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  Sodium, 7 Day Follow-up | 139.2 (2.27) | 138.5 (2.26)
  Sodium, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  Sodium, 28 Day Follow-up | 138.8 (1.93) | 138.8 (3.03)
  Calcium, Day 1: number analyzed (Participants) | 54 | 27
  Calcium, Day 1 | 2.264 (0.1523) | 2.251 (0.1169)
  Calcium, Day 4: number analyzed (Participants) | 44 | 24
  Calcium, Day 4 | 2.217 (0.1094) | 2.257 (0.0930)
  Calcium, Day 8: number analyzed (Participants) | 44 | 24
  Calcium, Day 8 | 2.267 (0.1055) | 2.273 (0.0719)
  Calcium, Day 11: number analyzed (Participants) | 40 | 23
  Calcium, Day 11 | 2.301 (0.1070) | 2.282 (0.0772)
  Calcium, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  Calcium, 7 Day Follow-up | 2.315 (0.1082) | 2.303 (0.0959)
  Calcium, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  Calcium, 28 Day Follow-up | 2.306 (0.1268) | 2.263 (0.0913)
  Potassium, Day 1: number analyzed (Participants) | 54 | 27
  Potassium, Day 1 | 4.18 (0.373) | 4.08 (0.297)
  Potassium, Day 4: number analyzed (Participants) | 44 | 24
  Potassium, Day 4 | 4.19 (0.400) | 4.11 (0.301)
  Potassium, Day 8: number analyzed (Participants) | 44 | 24
  Potassium, Day 8 | 4.18 (0.288) | 4.13 (0.303)
  Potassium, Day 11: number analyzed (Participants) | 40 | 23
  Potassium, Day 11 | 4.12 (0.280) | 4.04 (0.301)
  Potassium, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  Potassium, 7 Day Follow-up | 4.16 (0.331) | 4.06 (0.357)
  Potassium, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  Potassium, 28 Day Follow-up | 4.04 (0.307) | 4.13 (0.293)
  Chloride, Day 1: number analyzed (Participants) | 56 | 27
  Chloride, Day 1 | 102.3 (3.12) | 102.4 (3.55)
  Chloride, Day 4: number analyzed (Participants) | 45 | 25
  Chloride, Day 4 | 101.9 (3.71) | 103.0 (3.01)
  Chloride, Day 8: number analyzed (Participants) | 44 | 24
  Chloride, Day 8 | 102.9 (2.57) | 103.8 (2.95)
  Chloride, Day 11: number analyzed (Participants) | 40 | 23
  Chloride, Day 11 | 104.2 (2.69) | 102.7 (4.05)
  Chloride, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  Chloride, 7 Day Follow-up | 104.7 (2.14) | 102.6 (3.85)
  Chloride, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  Chloride, 28 Day Follow-up | 103.7 (2.60) | 103.7 (3.97)
  CO2 content/bicarbonate, Day 1: number analyzed (Participants) | 54 | 27
  CO2 content/bicarbonate, Day 1 | 21.7 (2.68) | 21.1 (2.43)
  CO2 content/bicarbonate, Day 4: number analyzed (Participants) | 44 | 24
  CO2 content/bicarbonate, Day 4 | 22.3 (2.51) | 23.0 (2.44)
  CO2 content/bicarbonate, Day 8: number analyzed (Participants) | 44 | 24
  CO2 content/bicarbonate, Day 8 | 22.2 (2.16) | 22.5 (2.08)
  CO2 content/bicarbonate, Day 11: number analyzed (Participants) | 40 | 23
  CO2 content/bicarbonate, Day 11 | 21.6 (2.20) | 22.8 (2.77)
  CO2 content/bicarbonate, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  CO2 content/bicarbonate, 7 Day Follow-up | 21.9 (2.31) | 22.0 (2.51)
  CO2 content/bicarbonate, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  CO2 content/bicarbonate, 28 Day Follow-up | 22.3 (2.05) | 21.5 (2.64)
  Urea/BUN, Day 1: number analyzed (Participants) | 55 | 27
  Urea/BUN, Day 1 | 4.90 (1.695) | 4.20 (1.137)
  Urea/BUN, Day 4: number analyzed (Participants) | 45 | 25
  Urea/BUN, Day 4 | 4.81 (1.383) | 4.48 (1.475)
  Urea/BUN, Day 8: number analyzed (Participants) | 44 | 24
  Urea/BUN, Day 8 | 4.47 (1.188) | 4.73 (1.452)
  Urea/BUN, Day 11: number analyzed (Participants) | 40 | 23
  Urea/BUN, Day 11 | 4.69 (1.381) | 4.87 (1.618)
  Urea/BUN, 7 Day Follow-up: number analyzed (Participants) | 45 | 24
  Urea/BUN, 7 Day Follow-up | 4.84 (1.665) | 5.00 (1.836)
  Urea/BUN, 28 Day Follow-up: number analyzed (Participants) | 40 | 23
  Urea/BUN, 28 Day Follow-up | 4.88 (1.526) | 4.85 (0.947)

6. Primary Outcome: Mean Clinical Chemistry Parameter of Estradiol at Indicated Time Point
Description: Blood samples were obtained for analysis of estradiol at Day 1.
Time Frame: Day 1
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picomole (pmol)/Liter
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 6 | 3
Picomole (pmol)/Liter | 261.8 (218.20) | 61.3 (22.37)

7. Primary Outcome: Mean Clinical Chemistry Parameter of High Sensitivity C-Reactive Protein at Indicated Time Points
Description: Blood samples were obtained for analysis of high sensitivity C-Reactive protein at Day 1, Day 2, Day 3, Day 4, Day 8, Day 11 and 7 Day Follow-up. Baseline value was defined as the assessment done on Day 1.
Time Frame: Up to Follow-up (7 Day Follow-up, Day 19)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mg/Liter
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
mg/Liter
  Day 1: number analyzed (Participants) | 55 | 27
  Day 1 | 38.39 (35.968) | 43.97 (42.829)
  Day 2: number analyzed (Participants) | 47 | 25
  Day 2 | 33.76 (36.759) | 40.72 (43.485)
  Day 3: number analyzed (Participants) | 46 | 26
  Day 3 | 27.13 (32.425) | 30.99 (42.930)
  Day 4: number analyzed (Participants) | 44 | 25
  Day 4 | 15.71 (23.564) | 21.82 (34.947)
  Day 8: number analyzed (Participants) | 43 | 24
  Day 8 | 6.87 (7.561) | 6.02 (5.280)
  Day 11: number analyzed (Participants) | 41 | 23
  Day 11 | 7.56 (9.711) | 4.74 (4.658)
  7 Day Follow-up: number analyzed (Participants) | 42 | 25
  7 Day Follow-up | 10.25 (16.299) | 7.29 (8.377)

8. Primary Outcome: Mean Hematology Parameters of Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, White Blood Cells (WBC) and Platelet Count at Indicated Time Points
Description: Blood samples were obtained for analysis of basophils, eosinophils, lymphocytes, monocytes, total neutrophils, WBC and platelet count at Day 1, Day 4, Day 8, Day 11, 7 Day Follow-up and 28 Day Follow-up. Baseline value was defined as the assessment done on Day 1.
Time Frame: Up to Follow-up (28 Day Follow-up, Day 40)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells/Liter
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Giga cells/Liter
  Basophils, Day 1: number analyzed (Participants) | 56 | 26
  Basophils, Day 1 | 0.027 (0.0146) | 0.035 (0.0272)
  Basophils, Day 4: number analyzed (Participants) | 44 | 25
  Basophils, Day 4 | 0.030 (0.0179) | 0.035 (0.0247)
  Basophils, Day 8: number analyzed (Participants) | 44 | 24
  Basophils, Day 8 | 0.027 (0.0125) | 0.035 (0.0343)
  Basophils, Day 11: number analyzed (Participants) | 40 | 23
  Basophils, Day 11 | 0.030 (0.0234) | 0.020 (0.0088)
  Basophils, 7 Day Follow-up: number analyzed (Participants) | 45 | 25
  Basophils, 7 Day Follow-up | 0.032 (0.0162) | 0.027 (0.0199)
  Basophils, 28 Day Follow-up: number analyzed (Participants) | 39 | 22
  Basophils, 28 Day Follow-up | 0.024 (0.0144) | 0.031 (0.0187)
  Eosinophils, Day 1: number analyzed (Participants) | 56 | 26
  Eosinophils, Day 1 | 0.149 (0.1116) | 0.140 (0.1022)
  Eosinophils, Day 4: number analyzed (Participants) | 44 | 25
  Eosinophils, Day 4 | 0.149 (0.1708) | 0.145 (0.1018)
  Eosinophils, Day 8: number analyzed (Participants) | 44 | 24
  Eosinophils, Day 8 | 0.165 (0.1347) | 0.155 (0.1016)
  Eosinophils, Day 11: number analyzed (Participants) | 40 | 23
  Eosinophils, Day 11 | 0.175 (0.1534) | 0.168 (0.1155)
  Eosinophils, 7 Day Follow-up: number analyzed (Participants) | 45 | 25
  Eosinophils, 7 Day Follow-up | 0.151 (0.0870) | 0.128 (0.0947)
  Eosinophils, 28 Day Follow-up: number analyzed (Participants) | 39 | 22
  Eosinophils, 28 Day Follow-up | 0.141 (0.1060) | 0.150 (0.0959)
  Monocytes, Day 1: number analyzed (Participants) | 56 | 26
  Monocytes, Day 1 | 0.432 (0.2097) | 0.517 (0.2131)
  Monocytes, Day 4: number analyzed (Participants) | 44 | 25
  Monocytes, Day 4 | 0.354 (0.1352) | 0.408 (0.2819)
  Monocytes, Day 8: number analyzed (Participants) | 44 | 24
  Monocytes, Day 8 | 0.370 (0.1265) | 0.388 (0.1826)
  Monocytes, Day 11: number analyzed (Participants) | 40 | 23
  Monocytes, Day 11 | 0.320 (0.1475) | 0.420 (0.1800)
  Monocytes, 7 Day Follow-up: number analyzed (Participants) | 45 | 25
  Monocytes, 7 Day Follow-up | 0.345 (0.1544) | 0.410 (0.1677)
  Monocytes, 28 Day Follow-up: number analyzed (Participants) | 39 | 22
  Monocytes, 28 Day Follow-up | 0.384 (0.1502) | 0.471 (0.2175)
  Total neutrophils, Day 1: number analyzed (Participants) | 56 | 26
  Total neutrophils, Day 1 | 6.533 (3.0198) | 7.231 (2.4074)
  Total neutrophils, Day 4: number analyzed (Participants) | 44 | 25
  Total neutrophils, Day 4 | 4.757 (2.1470) | 4.984 (2.0237)
  Total neutrophils, Day 8: number analyzed (Participants) | 44 | 24
  Total neutrophils, Day 8 | 4.371 (1.6688) | 4.780 (2.6362)
  Total neutrophils, Day 11: number analyzed (Participants) | 40 | 23
  Total neutrophils, Day 11 | 4.495 (2.0516) | 4.524 (1.7753)
  Total neutrophils, 7 Day Follow-up: number analyzed (Participants) | 45 | 25
  Total neutrophils, 7 Day Follow-up | 4.111 (1.5873) | 4.821 (2.0453)
  Total neutrophils, 28 Day Follow-up: number analyzed (Participants) | 39 | 22
  Total neutrophils, 28 Day Follow-up | 4.709 (1.9470) | 5.496 (2.9618)
  WBC count, Day 1: number analyzed (Participants) | 56 | 26
  WBC count, Day 1 | 9.15 (3.420) | 9.87 (2.673)
  WBC count, Day 4: number analyzed (Participants) | 44 | 25
  WBC count, Day 4 | 7.35 (2.551) | 7.54 (2.462)
  WBC count, Day 8: number analyzed (Participants) | 44 | 24
  WBC count, Day 8 | 6.82 (1.997) | 7.30 (2.895)
  WBC count, Day 11: number analyzed (Participants) | 40 | 23
  WBC count, Day 11 | 6.77 (2.209) | 7.06 (2.172)
  WBC count, 7 Day Follow-up: number analyzed (Participants) | 45 | 25
  WBC count, 7 Day Follow-up | 6.44 (2.077) | 7.48 (2.432)
  WBC count, 28 Day Follow-up: number analyzed (Participants) | 39 | 22
  WBC count, 28 Day Follow-up | 7.16 (2.415) | 8.10 (3.268)
  Platelet count, Day 1: number analyzed (Participants) | 55 | 25
  Platelet count, Day 1 | 285.5 (91.48) | 255.0 (72.48)
  Platelet count, Day 4: number analyzed (Participants) | 42 | 25
  Platelet count, Day 4 | 296.5 (93.96) | 273.2 (74.68)
  Platelet count, Day 8: number analyzed (Participants) | 44 | 24
  Platelet count, Day 8 | 293.0 (79.28) | 268.3 (56.90)
  Platelet count, Day 11: number analyzed (Participants) | 40 | 22
  Platelet count, Day 11 | 280.2 (78.24) | 253.9 (62.44)
  Platelet count, 7 Day Follow-up: number analyzed (Participants) | 45 | 25
  Platelet count, 7 Day Follow-up | 264.0 (71.40) | 249.8 (58.68)
  Platelet count, 28 Day Follow-up: number analyzed (Participants) | 38 | 22
  Platelet count, 28 Day Follow-up | 279.3 (74.61) | 240.5 (69.81)
  Lymphocytes, Day 1: number analyzed (Participants) | 56 | 26
  Lymphocytes, Day 1 | 2.012 (0.7487) | 1.947 (0.6455)
  Lymphocytes, Day 4: number analyzed (Participants) | 44 | 25
  Lymphocytes, Day 4 | 2.057 (0.8168) | 1.968 (0.6718)
  Lymphocytes, Day 8: number analyzed (Participants) | 44 | 24
  Lymphocytes, Day 8 | 1.890 (0.7039) | 1.941 (0.7312)
  Lymphocytes, Day 11: number analyzed (Participants) | 40 | 23
  Lymphocytes, Day 11 | 1.749 (0.6990) | 1.925 (0.6202)
  Lymphocytes, 7 Day Follow-up: number analyzed (Participants) | 45 | 25
  Lymphocytes, 7 Day Follow-up | 1.806 (0.7018) | 2.091 (0.8427)
  Lymphocytes, 28 Day Follow-up: number analyzed (Participants) | 39 | 22
  Lymphocytes, 28 Day Follow-up | 1.907 (0.7745) | 1.955 (0.4947)

9. Primary Outcome: Mean Hematology Parameter of Mean Corpuscle Volume (MCV) at Indicated Time Points
Description: Blood samples were obtained for analysis of MCV at Day 1, Day 4, Day 8, Day 11, 7 Day Follow-up and 28 Day Follow-up. Baseline value was defined as the assessment done on Day 1.
Time Frame: Up to Follow-up (28 Day Follow-up, Day 40)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Groups:
- GSK1322322 1500 mg: Participants received oral dose of GSK1322322 1500 mg as 3 tablets of 500 mg each, BID in the morning and evening for 10 days. Blinding was maintained by administration of matching placebo capsules to linezoid in the morning and evening. The study medication was taken with 240 mL of water or liquid.
- Linezolid 600 mg: Participants received oral dose of linezolid 600 mg tablet BID in the morning and evening for 10 days. Blinding was maintained by administration of matching placebo tablets to GSK1322322 in the morning and evening. The study medication was taken with 240 mL of water or liquid.
Arm/Group | GSK1322322 1500 mg | Linezolid 600 mg
Number analyzed (Participants) | 57 | 27
Femtoliter
  Day 1: number analyzed (Participants) | 56 | 26
  Day 1 | 90.5 (5.24) | 91.1 (8.53)
  Day 4: number analyzed (Participants) | 44 | 25
  Day 4 | 89.8 (5.52) | 91.6 (7.13)
  Day 8: number analyzed (Participants) | 44 | 24
  Day 8 | 89.4 (5.88) | 91.2 (7.01)
  Day 11: number analyzed (Participants) | 40 | 23
  Day 11 | 89.7 (5.38) | 90.7 (6.96)
  7 Day Follow-up: number analyzed (Participants) | 45 | 25
  7 Day Follow-up | 89.1 (4.91) | 91.5 (7.00)
  28 Day Follow-up: number analyzed (Participants) | 39 | 22
  28 Day Follow-up | 90.1 (5.60) | 91.3 (7.63)

10. Primary Outcome: Mean Hematology Parameter of Hemoglobin, Mean Corpuscle Hemoglobin Concentration (MCHC) at Indicated Time Points
Description: Blood samples were obtained for analysis of MCHC at Day 1, Day 4, Day 8, Day 11, 7 Day Follow-up and 28 Day Follow-up. Baseline value was defined as the assessment done on Day 1.
Time Frame: Up to Follow-up (28 Day Follow-up, Day 40)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Gram/Liter
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Gram/Liter
  Hemoglobin, Day 1: number analyzed (Participants) | 56 | 26
  Hemoglobin, Day 1 | 136.7 (15.67) | 134.2 (19.49)
  Hemoglobin, Day 4: number analyzed (Participants) | 44 | 25
  Hemoglobin, Day 4 | 132.9 (15.49) | 133.5 (18.44)
  Hemoglobin, Day 8: number analyzed (Participants) | 44 | 24
  Hemoglobin, Day 8 | 135.8 (16.47) | 134.0 (19.03)
  Hemoglobin, Day 11: number analyzed (Participants) | 40 | 23
  Hemoglobin, Day 11 | 135.9 (16.83) | 136.4 (19.04)
  Hemoglobin, 7 Day Follow-up: number analyzed (Participants) | 45 | 25
  Hemoglobin, 7 Day Follow-up | 137.7 (19.71) | 135.8 (19.08)
  Hemoglobin, 28 Day Follow-up: number analyzed (Participants) | 39 | 22
  Hemoglobin, 28 Day Follow-up | 139.6 (17.82) | 136.1 (18.35)
  MCHC, Day 1: number analyzed (Participants) | 56 | 26
  MCHC, Day 1 | 334.0 (8.73) | 331.9 (12.38)
  MCHC, Day 4: number analyzed (Participants) | 44 | 25
  MCHC, Day 4 | 335.1 (9.42) | 333.5 (15.25)
  MCHC, Day 8: number analyzed (Participants) | 44 | 24
  MCHC, Day 8 | 336.6 (8.73) | 335.7 (12.60)
  MCHC, Day 11: number analyzed (Participants) | 40 | 23
  MCHC, Day 11 | 335.5 (7.73) | 336.4 (14.24)
  MCHC, 7 Day Follow-up: number analyzed (Participants) | 45 | 25
  MCHC, 7 Day Follow-up | 337.8 (7.39) | 335.4 (10.67)
  MCHC, 28 Day Follow-up: number analyzed (Participants) | 39 | 22
  MCHC, 28 Day Follow-up | 336.1 (8.53) | 334.3 (11.80)

11. Primary Outcome: Mean Hematology Parameter of Mean Corpuscle Hemoglobin (MCH) at Indicated Time Points
Description: Blood samples were obtained for analysis of MCH at Day 1, Day 4, Day 8, Day 11, 7 Day Follow-up and 28 Day Follow-up. Baseline value was defined as the assessment done on Day 1.
Time Frame: Up to Follow-up (28 Day Follow-up, Day 40)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Picogram
  Day 1: number analyzed (Participants) | 56 | 26
  Day 1 | 30.22 (1.970) | 30.24 (3.284)
  Day 4: number analyzed (Participants) | 44 | 25
  Day 4 | 30.08 (2.169) | 30.58 (2.957)
  Day 8: number analyzed (Participants) | 44 | 24
  Day 8 | 30.10 (2.165) | 30.63 (2.970)
  Day 11: number analyzed (Participants) | 40 | 23
  Day 11 | 30.06 (2.107) | 30.59 (3.014)
  7 Day Follow-up: number analyzed (Participants) | 45 | 25
  7 Day Follow-up | 30.14 (2.021) | 30.71 (2.845)
  28 Day Follow-up: number analyzed (Participants) | 39 | 22
  28 Day Follow-up | 30.26 (2.070) | 30.56 (3.002)

12. Primary Outcome: Mean Hematology Parameter of Red Blood Cell (RBC) Count and Reticulocyte Count at Indicated Time Points
Description: Blood samples were obtained for analysis of RBC count and reticulocyte at Day 1, Day 4, Day 8, Day 11, 7 Day Follow-up and 28 Day Follow-up. Baseline value was defined as the assessment done on Day 1.
Time Frame: Up to Follow-up (28 Day Follow-up, Day 40)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Trillion cells (TI)/Liter
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Trillion cells (TI)/Liter
  RBC count, Day 1: number analyzed (Participants) | 56 | 26
  RBC count, Day 1 | 4.53 (0.413) | 4.43 (0.397)
  RBC count, Day 4: number analyzed (Participants) | 44 | 25
  RBC count, Day 4 | 4.43 (0.370) | 4.36 (0.454)
  RBC count, Day 8: number analyzed (Participants) | 44 | 24
  RBC count, Day 8 | 4.52 (0.430) | 4.37 (0.389)
  RBC count, Day 11: number analyzed (Participants) | 40 | 23
  RBC count, Day 11 | 4.52 (0.410) | 4.46 (0.436)
  RBC count, 7 Day Follow-up: number analyzed (Participants) | 45 | 25
  RBC count, 7 Day Follow-up | 4.56 (0.489) | 4.42 (0.457)
  RBC count, 28 Day Follow-up: number analyzed (Participants) | 39 | 22
  RBC count, 28 Day Follow-up | 4.61 (0.430) | 4.44 (0.376)
  Reticulocytes, Day 1: number analyzed (Participants) | 56 | 25
  Reticulocytes, Day 1 | 0.07 (0.032) | 0.06 (0.021)
  Reticulocytes, Day 4: number analyzed (Participants) | 44 | 25
  Reticulocytes, Day 4 | 0.06 (0.024) | 0.05 (0.020)
  Reticulocytes, Day 8: number analyzed (Participants) | 44 | 24
  Reticulocytes, Day 8 | 0.07 (0.026) | 0.05 (0.023)
  Reticulocytes, Day 11: number analyzed (Participants) | 40 | 23
  Reticulocytes, Day 11 | 0.07 (0.031) | 0.07 (0.025)
  Reticulocytes, 7 Day Follow-up: number analyzed (Participants) | 45 | 25
  Reticulocytes, 7 Day Follow-up | 0.06 (0.029) | 0.08 (0.027)
  Reticulocytes, 28 Day Follow-up: number analyzed (Participants) | 39 | 22
  Reticulocytes, 28 Day Follow-up | 0.07 (0.031) | 0.06 (0.023)

13. Primary Outcome: Mean Vital Sign Value of Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Indicated Time Points
Description: Vital sign assessments were conducted at Day 1 (pre-dose), Day 2 (pre-dose), Day 3 (pre-dose), Day 4 (4-12 hours post-dose), Day 8 (pre-dose) and Day 11. The assessments were made with the participant in a semi-supine position, having rested in that position for at least 10 minutes beforehand. Three BP measurements were taken at pre-dose on Day 1. The mean value recorded at pre-dose was classified as Baseline. Single BP was obtained at all other time points during the study.
Time Frame: Up to Day 11
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Millimeters of mercury (mmHg)
  DBP, Day 1 | 78.1 (10.39) | 74.5 (10.46)
  DBP, Day 2: number analyzed (Participants) | 52 | 25
  DBP, Day 2 | 76.0 (10.81) | 76.7 (9.70)
  DBP, Day 3: number analyzed (Participants) | 49 | 26
  DBP, Day 3 | 73.6 (10.92) | 77.3 (11.01)
  DBP, Day 4: number analyzed (Participants) | 46 | 25
  DBP, Day 4 | 69.7 (9.63) | 76.8 (12.02)
  DBP, Day 8: number analyzed (Participants) | 44 | 24
  DBP, Day 8 | 73.5 (10.77) | 72.1 (11.23)
  DBP, Day 11: number analyzed (Participants) | 41 | 24
  DBP, Day 11 | 73.6 (9.75) | 72.8 (10.97)
  SBP, Day 1 | 125.6 (14.21) | 123.1 (12.72)
  SBP, Day 2: number analyzed (Participants) | 52 | 25
  SBP, Day 2 | 119.2 (13.78) | 125.1 (12.74)
  SBP, Day 3: number analyzed (Participants) | 49 | 26
  SBP, Day 3 | 120.0 (14.52) | 126.9 (15.96)
  SBP, Day 4: number analyzed (Participants) | 46 | 25
  SBP, Day 4 | 119.3 (13.56) | 126.1 (14.83)
  SBP, Day 8: number analyzed (Participants) | 44 | 24
  SBP, Day 8 | 122.7 (14.78) | 121.2 (16.02)
  SBP, Day 11: number analyzed (Participants) | 41 | 24
  SBP, Day 11 | 122.0 (14.53) | 120.4 (13.25)

14. Primary Outcome: Mean Vital Sign Value of Heart Rate (HR) at Indicated Time Points
Description: Vital sign assessments were conducted at Day 1 (pre-dose), Day 2 (pre-dose), Day 3 (pre-dose), Day 4 (4-12 hours post-dose), Day 8 (pre-dose) and Day 11. The assessments were made with the participant in a semi-supine position, having rested in that position for at least 10 minutes beforehand. Three HR measurements were taken at pre-dose on Day 1. The mean value recorded at pre-dose was classified as Baseline. Single HR was obtained at all other time points during the study.
Time Frame: Up to Day 11
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Beats per minute
  Day 1 | 74.9 (13.75) | 73.9 (14.11)
  Day 2: number analyzed (Participants) | 52 | 25
  Day 2 | 81.2 (14.54) | 76.2 (12.80)
  Day 3: number analyzed (Participants) | 49 | 26
  Day 3 | 77.6 (12.81) | 76.1 (11.70)
  Day 4: number analyzed (Participants) | 46 | 25
  Day 4 | 71.9 (11.21) | 74.6 (17.08)
  Day 8: number analyzed (Participants) | 44 | 24
  Day 8 | 69.9 (10.52) | 69.2 (12.07)
  Day 11: number analyzed (Participants) | 41 | 24
  Day 11 | 70.9 (12.86) | 74.0 (12.22)

15. Primary Outcome: Mean Vital Sign Value of Respiratory Rate (RR) at Indicated Time Points
Description: Vital sign assessments were conducted at Day 1 (pre-dose), Day 2 (pre-dose), Day 3 (pre-dose), Day 4 (4-12 hours post-dose), Day 8 (pre-dose) and Day 11. The assessments were made with the participant in a semi-supine position, having rested in that position for at least 10 minutes beforehand. Three RR measurements were taken at pre-dose on Day 1. The mean value recorded at pre-dose was classified as Baseline. Single RR was obtained at all other time points during the study.
Time Frame: Up to Day 11
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Breaths per minute
  Day 1 | 17.1 (1.95) | 17.9 (1.70)
  Day 2: number analyzed (Participants) | 52 | 25
  Day 2 | 17.3 (1.78) | 17.4 (1.98)
  Day 3: number analyzed (Participants) | 49 | 26
  Day 3 | 17.4 (2.08) | 17.3 (1.85)
  Day 4: number analyzed (Participants) | 46 | 25
  Day 4 | 17.3 (1.92) | 17.4 (1.85)
  Day 8: number analyzed (Participants) | 44 | 24
  Day 8 | 17.1 (1.66) | 17.2 (1.76)
  Day 11: number analyzed (Participants) | 41 | 24
  Day 11 | 17.6 (2.20) | 16.8 (1.96)

16. Primary Outcome: Mean Change From Baseline in SBP and DBP at Indicated Time Points
Description: Vital sign assessments were conducted at Day 1 (pre-dose), Day 2 (pre-dose), Day 3 (pre-dose), Day 4 (4-12 hours post-dose), Day 8 (pre-dose) and Day 11. The assessments were made with the participant in a semi-supine position, having rested in that position for at least 10 minutes beforehand. Three BP measurements were taken at pre-dose on Day 1. The mean value recorded at pre-dose was classified as Baseline. Single BP was obtained at all other time points during the study. The change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 2, Day 3, Day 4, Day 8 and Day 11) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to missing as well.
Time Frame: Day 1 (Baseline) up to Day 11
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
mmHg
  SBP, Day 2: number analyzed (Participants) | 52 | 25
  SBP, Day 2 | -6.5 (12.23) | 1.6 (15.35)
  SBP, Day 3: number analyzed (Participants) | 49 | 26
  SBP, Day 3 | -5.2 (11.24) | 3.7 (18.64)
  SBP, Day 4: number analyzed (Participants) | 46 | 25
  SBP, Day 4 | -6.5 (11.31) | 3.1 (15.21)
  SBP, Day 8: number analyzed (Participants) | 44 | 24
  SBP, Day 8 | -2.5 (12.23) | -2.7 (13.95)
  SBP, Day 11: number analyzed (Participants) | 41 | 24
  SBP, Day 11 | -2.7 (12.70) | -2.6 (15.44)
  DBP, Day 2: number analyzed (Participants) | 52 | 25
  DBP, Day 2 | -2.6 (8.64) | 1.8 (6.46)
  DBP, Day 3: number analyzed (Participants) | 49 | 26
  DBP, Day 3 | -4.8 (8.64) | 2.7 (13.59)
  DBP, Day 4: number analyzed (Participants) | 46 | 25
  DBP, Day 4 | -8.7 (9.02) | 2.5 (12.10)
  DBP, Day 8: number analyzed (Participants) | 44 | 24
  DBP, Day 8 | -4.7 (9.92) | -2.8 (11.00)
  DBP, Day 11: number analyzed (Participants) | 41 | 24
  DBP, Day 11 | -4.4 (7.61) | -1.7 (9.53)

17. Primary Outcome: Mean Change From Baseline in HR at Indicated Time Points
Description: Vital sign assessments were conducted at Day 1 (pre-dose), Day 2 (pre-dose), Day 3 (pre-dose), Day 4 (4-12 hours post-dose), Day 8 (pre-dose) and Day 11. The assessments were made with the participant in a semi-supine position, having rested in that position for at least 10 minutes beforehand. Three HR measurements were taken at pre-dose on Day 1. The mean value recorded at pre-dose was classified as Baseline. Single HR was obtained at all other time points during the study. The change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 2, Day 3, Day 4, Day 8 and Day 11) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to missing as well.
Time Frame: Day 1 (Baseline) up to Day 11
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Beats per minute
  Day 2: number analyzed (Participants) | 52 | 25
  Day 2 | 6.5 (13.74) | 3.7 (11.93)
  Day 3: number analyzed (Participants) | 49 | 26
  Day 3 | 2.2 (11.47) | 4.0 (11.48)
  Day 4: number analyzed (Participants) | 46 | 25
  Day 4 | -1.4 (10.28) | 2.5 (19.57)
  Day 8: number analyzed (Participants) | 44 | 24
  Day 8 | -3.0 (10.98) | -2.7 (12.05)
  Day 11: number analyzed (Participants) | 41 | 24
  Day 11 | -2.5 (12.07) | 1.7 (12.28)

18. Primary Outcome: Mean Change From Baseline in RR at Indicated Time Points
Description: Vital sign assessments were conducted at Day 1 (pre-dose), Day 2 (pre-dose), Day 3 (pre-dose), Day 4 (4-12 hours post-dose), Day 8 (pre-dose) and Day 11. The assessments were made with the participant in a semi-supine position, having rested in that position for at least 10 minutes beforehand. Three RR measurements were taken at pre-dose on Day 1. The mean value recorded at pre-dose was classified as Baseline. Single RR was obtained at all other time points during the study. The change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 2, Day 3, Day 4, Day 8 and Day 11) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to missing as well.
Time Frame: Day 1 (Baseline) up to Day 11
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Breaths per minute
  Day 2: number analyzed (Participants) | 52 | 25
  Day 2 | 0.4 (1.80) | -0.7 (2.07)
  Day 3: number analyzed (Participants) | 49 | 26
  Day 3 | 0.5 (2.41) | -0.7 (1.43)
  Day 4: number analyzed (Participants) | 46 | 25
  Day 4 | 0.4 (2.35) | -0.6 (2.14)
  Day 8: number analyzed (Participants) | 44 | 24
  Day 8 | 0.2 (1.98) | -0.8 (1.75)
  Day 11: number analyzed (Participants) | 41 | 24
  Day 11 | 0.6 (2.11) | -1.2 (1.89)

19. Primary Outcome: Mean Electrocardiogram (ECG) Values at Indicated Time Points
Description: 12-lead ECGs were obtained during the study using an ECG machine that automatically calculated the heart rate and measured PR, QRS, RR, QT, and QTc intervals. It was performed with the participant in a semi-supine position having rested in that position for at least 10 minutes beforehand. Three measurements were taken at pre-dose on Day 1 at least 5 minutes apart. The mean PR interval, RR interval, QRS duration, uncorrected QT interval (UncQT) and QTcB (QT corrected by Bazett's formula) and QTcF (corrected by Friedericia's formula) was calculated from automated ECG readings. The assessments were done at Day 1 (pre-dose, 0.25-1.5 hours post-initial dose and 1.5-3 hours post-initial dose), Day 4 (4-12 hours post-morning dose), Day 8 (pre-morning dose) and Day 11 (0 hour). The mean value recorded pre-dose on Day 1 was classified as Baseline.
Time Frame: Up to Day 11
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millisecond (msec)
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Millisecond (msec)
  PR interval, Day 1, mean pre-dose | 158.0 (15.88) | 155.0 (20.17)
  PR interval, Day 1, 0.25-1.5 h post-dose | 157.0 (15.80) | 159.2 (22.72)
  PR interval, Day 1,1.5-3 h post-dose: number analyzed (Participants) | 56 | 26
  PR interval, Day 1,1.5-3 h post-dose | 158.5 (17.07) | 157.2 (23.87)
  PR interval, Day 4, 4-12 h post-dose: number analyzed (Participants) | 46 | 25
  PR interval, Day 4, 4-12 h post-dose | 165.8 (18.35) | 159.2 (21.39)
  PR interval, Day 8, pre morning dose: number analyzed (Participants) | 44 | 23
  PR interval, Day 8, pre morning dose | 167.4 (16.52) | 158.1 (23.98)
  PR interval, Day 11, 0 h: number analyzed (Participants) | 41 | 24
  PR interval, Day 11, 0 h | 158.6 (19.72) | 159.3 (19.37)
  QRS duration, Day 1, mean pre-dose | 94.0 (8.94) | 95.9 (6.67)
  QRS duration, Day 1, 0.25-1.5 h post-dose | 93.9 (9.19) | 97.1 (6.70)
  QRS duration, Day 1,1.5-3 h post-dose: number analyzed (Participants) | 56 | 26
  QRS duration, Day 1,1.5-3 h post-dose | 95.7 (8.76) | 96.1 (8.40)
  QRS duration, Day 4, 4-12 h post-dose: number analyzed (Participants) | 46 | 25
  QRS duration, Day 4, 4-12 h post-dose | 95.7 (8.91) | 93.7 (6.76)
  QRS duration, Day 8, pre morning dose: number analyzed (Participants) | 44 | 23
  QRS duration, Day 8, pre morning dose | 95.5 (10.07) | 95.3 (8.81)
  QRS duration, Day 11, 0 h: number analyzed (Participants) | 41 | 24
  QRS duration, Day 11, 0 h | 95.2 (8.41) | 96.2 (8.22)
  UncQT interval, Day 1, mean pre-dose | 376.7 (36.76) | 378.2 (39.50)
  UncQT interval, Day 1, 0.25-1.5 h post-dose | 370.8 (35.79) | 375.1 (28.51)
  UncQT interval, Day 1,1.5-3 h post-dose: number analyzed (Participants) | 56 | 26
  UncQT interval, Day 1,1.5-3 h post-dose | 370.3 (36.01) | 374.0 (25.42)
  UncQT interval, Day 4, 4-12 h post-dose: number analyzed (Participants) | 46 | 24
  UncQT interval, Day 4, 4-12 h post-dose | 392.6 (32.26) | 378.4 (37.77)
  UncQT interval, Day 8, pre morning dose: number analyzed (Participants) | 44 | 22
  UncQT interval, Day 8, pre morning dose | 397.1 (31.64) | 390.3 (27.18)
  UncQT interval, Day 11, 0 h: number analyzed (Participants) | 41 | 24
  UncQT interval, Day 11, 0 h | 385.3 (32.05) | 382.2 (41.47)
  QTcB interval, Day 1, mean pre-dose | 416.0 (26.09) | 411.6 (28.57)
  QTcB interval, Day 1, 0.25-1.5 h post-dose | 421.1 (22.91) | 407.9 (28.74)
  QTcB interval, Day 1,1.5-3 h post-dose: number analyzed (Participants) | 56 | 26
  QTcB interval, Day 1,1.5-3 h post-dose | 424.1 (24.89) | 412.7 (25.40)
  QTcB interval, Day 4, 4-12 h post-dose: number analyzed (Participants) | 46 | 24
  QTcB interval, Day 4, 4-12 h post-dose | 422.9 (23.65) | 413.2 (22.61)
  QTcB interval, Day 8, pre morning dose: number analyzed (Participants) | 44 | 22
  QTcB interval, Day 8, pre morning dose | 420.1 (22.82) | 411.0 (26.94)
  QTcB interval, Day 11, 0 h: number analyzed (Participants) | 41 | 24
  QTcB interval, Day 11, 0 h | 414.5 (17.76) | 413.1 (22.21)
  QTcF interval, Day 1, mean pre-dose | 402.0 (24.04) | 399.7 (28.20)
  QTcF interval, Day 1, 0.25-1.5 h post-dose | 403.1 (22.51) | 396.3 (24.78)
  QTcF interval, Day 1,1.5-3 h post-dose: number analyzed (Participants) | 56 | 26
  QTcF interval, Day 1,1.5-3 h post-dose | 405.0 (24.14) | 399.2 (22.47)
  QTcF interval, Day 4, 4-12 h post-dose: number analyzed (Participants) | 46 | 24
  QTcF interval, Day 4, 4-12 h post-dose | 412.3 (22.76) | 400.9 (21.28)
  QTcF interval, Day 8, pre morning dose: number analyzed (Participants) | 44 | 22
  QTcF interval, Day 8, pre morning dose | 412.0 (21.87) | 403.7 (21.54)
  QTcF interval, Day 11, 0 h: number analyzed (Participants) | 41 | 24
  QTcF interval, Day 11, 0 h | 404.1 (16.95) | 402.0 (24.27)
  RR interval, Day 1, mean pre-dose | 832.9 (173.04) | 854.6 (150.70)
  RR interval, Day 1, 0.25-1.5 h post-dose | 783.8 (148.25) | 855.0 (126.77)
  RR interval, Day 1,1.5-3 h post-dose: number analyzed (Participants) | 56 | 26
  RR interval, Day 1,1.5-3 h post-dose | 770.7 (149.27) | 825.8 (101.01)
  RR interval, Day 4, 4-12 h post-dose: number analyzed (Participants) | 46 | 25
  RR interval, Day 4, 4-12 h post-dose | 868.7 (133.65) | 860.7 (185.66)
  RR interval, Day 8, pre morning dose: number analyzed (Participants) | 44 | 23
  RR interval, Day 8, pre morning dose | 900.4 (134.96) | 918.6 (150.00)
  RR interval, Day 11, 0 h: number analyzed (Participants) | 41 | 24
  RR interval, Day 11, 0 h | 873.4 (155.04) | 865.0 (170.76)

20. Primary Outcome: Mean Change From Baseline in ECG Values at Indicated Time Points
Description: 12-lead ECGs were obtained during the study using an ECG machine that automatically calculated the heart rate and measured PR, QRS, RR, QT, and QTc intervals. It was performed with the participant in a semi-supine position having rested in that position for at least 10 minutes beforehand. Three measurements were taken at pre-dose on Day 1 at least 5 minutes apart. The mean PR interval, RR interval, QRS duration, uncorrected QT interval (UncQT) and QTcB (QT corrected by Bazett's formula) and QTcF (corrected by Friedericia's formula) was calculated from automated ECG readings. The assessments were done at Day 1 (pre-dose, 0.25-1.5 hours post-initial dose and 1.5-3 hours post-initial dose), Day 4 (4-12 hours post-morning dose), Day 8 (pre-morning dose) and Day 11 (0 hour). Mean value recorded pre-dose on Day 1 was classified as Baseline. Change from Baseline was calculated by subtracting the Baseline value from individual post-Baseline (Day 1 post-dose, Day 4, Day 8 and Day 11) values.
Time Frame: Day 1 (pre-dose, Baseline) up to Day 11
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
msec
  PR interval, Day 1, 0.25-1.5 h post dose | -1.0 (9.64) | 4.2 (12.88)
  PR interval, Day 1, 1.5-3 h post dose: number analyzed (Participants) | 56 | 26
  PR interval, Day 1, 1.5-3 h post dose | 0.4 (12.09) | 1.3 (11.79)
  PR interval, Day 4, 4-12 h post dose: number analyzed (Participants) | 46 | 25
  PR interval, Day 4, 4-12 h post dose | 6.3 (11.03) | 2.2 (11.75)
  PR interval, Day 8, pre morning dose: number analyzed (Participants) | 44 | 23
  PR interval, Day 8, pre morning dose | 7.1 (12.08) | -0.0 (13.79)
  PR interval, Day 11, 0 h: number analyzed (Participants) | 41 | 24
  PR interval, Day 11, 0 h | -1.2 (13.86) | 1.5 (14.27)
  QRS duration, Day 1, 0.25-1.5 h post dose | -0.2 (6.32) | 1.2 (5.52)
  QRS duration, Day 1, 1.5-3 h post dose: number analyzed (Participants) | 56 | 26
  QRS duration, Day 1, 1.5-3 h post dose | 1.6 (5.85) | 0.3 (6.84)
  QRS duration, Day 4, 4-12 h post dose: number analyzed (Participants) | 46 | 25
  QRS duration, Day 4, 4-12 h post dose | 1.6 (5.25) | -2.2 (7.28)
  QRS duration, Day 8, pre morning dose: number analyzed (Participants) | 44 | 23
  QRS duration, Day 8, pre morning dose | 1.0 (6.54) | -0.2 (8.18)
  QRS duration, Day 11, 0 h: number analyzed (Participants) | 41 | 24
  QRS duration, Day 11, 0 h | 1.2 (7.19) | -0.2 (7.50)
  UncQT interval, Day 1, 0.25-1.5 h post dose | -6.0 (18.66) | -3.1 (15.70)
  UncQT interval, Day 1, 1.5-3 h post dose: number analyzed (Participants) | 56 | 26
  UncQT interval, Day 1, 1.5-3 h post dose | -7.1 (19.33) | -7.2 (20.09)
  UncQT interval, Day 4, 4-12 h post dose: number analyzed (Participants) | 46 | 24
  UncQT interval, Day 4, 4-12 h post dose | 14.1 (24.16) | 0.5 (36.55)
  UncQT interval, Day 8, pre morning dose: number analyzed (Participants) | 44 | 22
  UncQT interval, Day 8, pre morning dose | 17.6 (29.12) | 10.5 (26.68)
  UncQT interval, Day 11, 0 h: number analyzed (Participants) | 41 | 24
  UncQT interval, Day 11, 0 h | 8.2 (30.04) | 1.5 (29.88)
  QTcB interval, Day 1, 0.25-1.5 h post dose | 5.1 (18.67) | -3.8 (13.50)
  QTcB interval, Day 1, 1.5-3 h post dose: number analyzed (Participants) | 56 | 26
  QTcB interval, Day 1, 1.5-3 h post dose | 8.5 (16.86) | 1.9 (17.59)
  QTcB interval, Day 4, 4-12 h post dose: number analyzed (Participants) | 46 | 24
  QTcB interval, Day 4, 4-12 h post dose | 8.4 (21.55) | 7.3 (16.70)
  QTcB interval, Day 8, pre morning dose: number analyzed (Participants) | 44 | 22
  QTcB interval, Day 8, pre morning dose | 5.4 (23.19) | 3.3 (21.13)
  QTcB interval, Day 11, 0 h: number analyzed (Participants) | 41 | 24
  QTcB interval, Day 11, 0 h | 0.0 (19.45) | 3.0 (20.16)
  QTcF interval, Day 1, 0.25-1.5 h post dose | 1.1 (14.99) | -3.4 (10.86)
  QTcF interval, Day 1, 1.5-3 h post dose: number analyzed (Participants) | 56 | 26
  QTcF interval, Day 1, 1.5-3 h post dose | 3.0 (13.39) | -1.2 (14.74)
  QTcF interval, Day 4, 4-12 h post dose: number analyzed (Participants) | 46 | 24
  QTcF interval, Day 4, 4-12 h post dose | 10.6 (16.68) | 4.9 (16.57)
  QTcF interval, Day 8, pre morning dose: number analyzed (Participants) | 44 | 22
  QTcF interval, Day 8, pre morning dose | 9.8 (19.31) | 5.9 (17.99)
  QTcF interval, Day 11, 0 h: number analyzed (Participants) | 41 | 24
  QTcF interval, Day 11, 0 h | 2.9 (18.09) | 2.3 (18.28)
  RR interval, Day 1, 0.25-1.5 h post dose | -49.2 (108.01) | 0.4 (88.51)
  RR interval, Day 1, 1.5-3 h post dose: number analyzed (Participants) | 56 | 26
  RR interval, Day 1, 1.5-3 h post dose | -66.4 (104.58) | -43.0 (102.48)
  RR interval, Day 4, 4-12 h post dose: number analyzed (Participants) | 46 | 25
  RR interval, Day 4, 4-12 h post dose | 23.7 (143.89) | -12.2 (194.88)
  RR interval, Day 8, pre morning dose: number analyzed (Participants) | 44 | 23
  RR interval, Day 8, pre morning dose | 51.6 (160.59) | 44.6 (146.43)
  RR interval, Day 11, 0 h: number analyzed (Participants) | 41 | 24
  RR interval, Day 11, 0 h | 33.9 (142.01) | -5.1 (153.97)

21. Primary Outcome: Mean ECG Rhythms at Indicated Time Points
Description: 12-lead ECGs were obtained during the study using an ECG machine that automatically calculated the heart rhythm and measured PR, QRS, RR, QT, and QTc intervals. It was performed with the participant in a semi-supine position having rested in that position for at least 10 minutes beforehand. Three measurements were taken at pre-dose on Day 1 at least 5 minutes apart and the mean of the three measurements was calculated. The assessments were done at Day 1 (pre-dose, 0.25-1.5 hours post-initial dose and 1.5-3 hours post-initial dose), Day 4 (4-12 hours post-morning dose), Day 8 (pre-morning dose) and Day 11 (0 hour).
Time Frame: Up to Day 11
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Beats per minute
  Day 1, mean pre-dose | 75.0 (14.33) | 72.8 (15.01)
  Day 1, 0.25-1.5 h post-dose | 79.2 (14.34) | 72.0 (13.04)
  Day 1,1.5-3 h post-dose: number analyzed (Participants) | 56 | 26
  Day 1,1.5-3 h post-dose | 80.4 (14.22) | 73.7 (9.19)
  Day 4, 4-12 h post-dose: number analyzed (Participants) | 46 | 25
  Day 4, 4-12 h post-dose | 70.6 (10.67) | 73.0 (16.39)
  Day 8, pre-morning dose: number analyzed (Participants) | 44 | 23
  Day 8, pre-morning dose | 68.2 (10.37) | 67.2 (12.28)
  Day 11, 0 h: number analyzed (Participants) | 41 | 24
  Day 11, 0 h | 70.9 (13.15) | 72.0 (13.94)

22. Primary Outcome: Mean Change From Baseline in ECG Rhythms at Indicated Time Points
Description: 12-lead ECGs were obtained during the study using an ECG machine that automatically calculated the heart rhythm and measured PR, QRS, RR, QT, and QTc intervals. It was performed with the participant in a semi-supine position having rested in that position for at least 10 minutes beforehand. Three measurements were taken at pre-dose on Day 1 at least 5 minutes apart and the mean of the three measurements was calculated. The assessments were done at Day 1 (pre-dose, 0.25-1.5 hours post-initial dose and 1.5-3 hours post-initial dose), Day 4 (4-12 hours post-morning dose), Day 8 (pre-morning dose) and Day 11 (0 hour). The value recorded pre-dose on Day 1 was the Baseline. The change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 1 post-dose, Day 4, Day 8 and Day 11) values.
Time Frame: Day 1 (pre-dose, Baseline) up to Day 11
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Beats per minute
  Day 1, 0.25-1.5 h post-dose | 4.2 (8.69) | -0.9 (6.29)
  Day 1, 1.5-3 h post-dose: number analyzed (Participants) | 56 | 26
  Day 1, 1.5-3 h post-dose | 5.9 (9.23) | 2.9 (8.35)
  Day 4, 4-12 h post-dose: number analyzed (Participants) | 46 | 25
  Day 4, 4-12 h post-dose | -3.1 (11.37) | 2.4 (16.48)
  Day 8, pre morning dose: number analyzed (Participants) | 44 | 23
  Day 8, pre morning dose | -5.2 (12.40) | -3.5 (10.12)
  Day 11, 0 h: number analyzed (Participants) | 41 | 24
  Day 11, 0 h | -3.2 (11.94) | 1.1 (11.39)

23. Primary Outcome: Number of Participants With Abnormal Transition From Baseline in Clinical Chemistry Values Relative to Normal Range
Description: The parameters of clinical chemistry included albumin, total protein, ALT, ALP, AST, GGT, LDH and creatine kinase, creatinine, uric acid, direct bilirubin, total bilirubin, glucose, sodium, calcium, potassium, chloride, CO2 content /bicarbonate and urea/BUN and high sensitivity C-Reactive protein. The assessments were done at Day 1, Day 4, Day 8, Day 11, 7 Day Follow-up and 28 Day Follow-up. Baseline was defined as the assessment done on Day 1 (pre-dose). Data is reported for number of participants with abnormal transition from Baseline 'to high' or 'to low' relative to normal range. Only those parameters for which at least one value of abnormal transition was reported are summarized.
Time Frame: Day 1 (pre-dose, Baseline) up Follow-up (28 Day Follow-up, Day 40)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Participants
  Day 2, C-Reactive protein, to high: number analyzed (Participants) | 48 | 25
  Day 2, C-Reactive protein, to high | 1 | 0
  Day 3, C-Reactive protein, to high: number analyzed (Participants) | 46 | 26
  Day 3, C-Reactive protein, to high | 1 | 0
  Day 4, ALT, to high: number analyzed (Participants) | 45 | 25
  Day 4, ALT, to high | 1 | 0
  Day 4, ALP, to high: number analyzed (Participants) | 45 | 25
  Day 4, ALP, to high | 1 | 0
  Day 4, AST, to high: number analyzed (Participants) | 44 | 24
  Day 4, AST, to high | 2 | 1
  Day 4, Calcium, to low: number analyzed (Participants) | 44 | 24
  Day 4, Calcium, to low | 6 | 0
  Day 4, CO2/bicarbonate, to low: number analyzed (Participants) | 44 | 24
  Day 4, CO2/bicarbonate, to low | 4 | 3
  Day 4, Chloride, to low: number analyzed (Participants) | 45 | 25
  Day 4, Chloride, to low | 1 | 0
  Day 4, Creatine kinase, to high: number analyzed (Participants) | 45 | 25
  Day 4, Creatine kinase, to high | 5 | 3
  Day 4, Creatinine, to low: number analyzed (Participants) | 45 | 25
  Day 4, Creatinine, to low | 2 | 2
  Day 4, GGT, to high: number analyzed (Participants) | 45 | 25
  Day 4, GGT, to high | 3 | 1
  Day 4, Glucose, to low: number analyzed (Participants) | 45 | 25
  Day 4, Glucose, to low | 2 | 0
  Day 4, Glucose, to high: number analyzed (Participants) | 45 | 25
  Day 4, Glucose, to high | 7 | 2
  Day 4, Potassium, to low: number analyzed (Participants) | 44 | 24
  Day 4, Potassium, to low | 1 | 0
  Day 4, Sodium, to low: number analyzed (Participants) | 45 | 25
  Day 4, Sodium, to low | 6 | 0
  Day 4, Total protein, to low: number analyzed (Participants) | 45 | 25
  Day 4, Total protein, to low | 1 | 1
  Day 4, Urea/BUN, to low: number analyzed (Participants) | 45 | 25
  Day 4, Urea/BUN, to low | 2 | 0
  Day 4, Urea/BUN, to high: number analyzed (Participants) | 45 | 25
  Day 4, Urea/BUN, to high | 0 | 1
  Day 4, Uric acid, to low: number analyzed (Participants) | 45 | 25
  Day 4, Uric acid, to low | 5 | 0
  Day 8, ALT, to high: number analyzed (Participants) | 44 | 24
  Day 8, ALT, to high | 1 | 2
  Day 8, Albumin, to low: number analyzed (Participants) | 44 | 24
  Day 8, Albumin, to low | 1 | 0
  Day 8, AST, to high: number analyzed (Participants) | 44 | 24
  Day 8, AST, to high | 4 | 2
  Day 8, Calcium, to low: number analyzed (Participants) | 44 | 24
  Day 8, Calcium, to low | 3 | 0
  Day 8, Chloride, to high: number analyzed (Participants) | 44 | 24
  Day 8, Chloride, to high | 1 | 0
  Day 8, Creatine kinase, to high: number analyzed (Participants) | 44 | 24
  Day 8, Creatine kinase, to high | 4 | 1
  Day 8, Creatinine, to low: number analyzed (Participants) | 44 | 24
  Day 8, Creatinine, to low | 4 | 1
  Day 8, GGT, to high: number analyzed (Participants) | 44 | 24
  Day 8, GGT, to high | 4 | 1
  Day 8, Glucose, to low: number analyzed (Participants) | 44 | 24
  Day 8, Glucose, to low | 1 | 1
  Day 8, Glucose, to high: number analyzed (Participants) | 44 | 24
  Day 8, Glucose, to high | 7 | 5
  Day 8, Sodium, to low: number analyzed (Participants) | 44 | 24
  Day 8, Sodium, to low | 1 | 1
  Day 8, Urea/BUN, to low: number analyzed (Participants) | 44 | 24
  Day 8, Urea/BUN, to low | 2 | 0
  Day 8, Uric acid, to low: number analyzed (Participants) | 44 | 24
  Day 8, Uric acid, to low | 2 | 0
  Day 11, ALT, to high: number analyzed (Participants) | 40 | 23
  Day 11, ALT, to high | 3 | 2
  Day 11, AST, to high: number analyzed (Participants) | 40 | 23
  Day 11, AST, to high | 5 | 2
  Day 11, Calcium, to low: number analyzed (Participants) | 40 | 23
  Day 11, Calcium, to low | 1 | 0
  Day 11, CO2/bicarbonate, to low: number analyzed (Participants) | 40 | 23
  Day 11, CO2/bicarbonate, to low | 5 | 2
  Day 11, Chloride, to low: number analyzed (Participants) | 40 | 23
  Day 11, Chloride, to low | 0 | 1
  Day 11, Chloride, to high: number analyzed (Participants) | 40 | 23
  Day 11, Chloride, to high | 1 | 1
  Day 11, Creatine kinase, to high: number analyzed (Participants) | 40 | 23
  Day 11, Creatine kinase, to high | 2 | 0
  Day 11, Creatinine, to low: number analyzed (Participants) | 40 | 23
  Day 11, Creatinine, to low | 2 | 2
  Day 11, GGT, to high: number analyzed (Participants) | 40 | 23
  Day 11, GGT, to high | 3 | 0
  Day 11, Glucose, to low: number analyzed (Participants) | 40 | 23
  Day 11, Glucose, to low | 3 | 0
  Day 11, Glucose, to high: number analyzed (Participants) | 40 | 23
  Day 11, Glucose, to high | 8 | 2
  Day 11, C-Reactive protein, to high: number analyzed (Participants) | 41 | 23
  Day 11, C-Reactive protein, to high | 1 | 1
  Day 11, Potassium, to low: number analyzed (Participants) | 40 | 23
  Day 11, Potassium, to low | 0 | 1
  Day 11, Sodium, to low: number analyzed (Participants) | 40 | 23
  Day 11, Sodium, to low | 0 | 1
  Day 11, Total protein, to high: number analyzed (Participants) | 40 | 23
  Day 11, Total protein, to high | 1 | 0
  Day 11, Urea/BUN, to low: number analyzed (Participants) | 40 | 23
  Day 11, Urea/BUN, to low | 2 | 0
  Day 11, Urea/BUN, to high: number analyzed (Participants) | 40 | 23
  Day 11, Urea/BUN, to high | 0 | 1
  Day 11, Uric acid, to low: number analyzed (Participants) | 40 | 23
  Day 11, Uric acid, to low | 0 | 1
  Day 11, Uric acid, to high: number analyzed (Participants) | 40 | 23
  Day 11, Uric acid, to high | 2 | 0
  7 Day Follow-up, ALT, to high: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, ALT, to high | 6 | 3
  7 Day Follow-up, AST, to high: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, AST, to high | 6 | 0
  7 Day Follow-up, Calcium, to low: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Calcium, to low | 1 | 0
  7 Day Follow-up, Calcium, to high: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Calcium, to high | 1 | 0
  7 Day Follow-up, CO2/bicarbonate, to low: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, CO2/bicarbonate, to low | 4 | 2
  7 Day Follow-up, Chloride, to low: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Chloride, to low | 0 | 1
  7 Day Follow-up, Chloride, to high: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Chloride, to high | 1 | 1
  7 Day Follow-up, Creatine kinase, to high: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Creatine kinase, to high | 4 | 3
  7 Day Follow-up, Creatinine, to low: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Creatinine, to low | 4 | 3
  7 Day Follow-up, Creatinine, to high: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Creatinine, to high | 0 | 1
  7 Day Follow-up, Direct bilirubin, to high: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Direct bilirubin, to high | 1 | 0
  7 Day Follow-up, GGT, to high: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, GGT, to high | 3 | 0
  7 Day Follow-up, Glucose, to high: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Glucose, to high | 4 | 2
  7 Day Follow-up, C-Reactive protein, to high: number analyzed (Participants) | 44 | 25
  7 Day Follow-up, C-Reactive protein, to high | 0 | 1
  7 Day Follow-up, Potassium, to low: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Potassium, to low | 1 | 1
  7 Day Follow-up, Sodium, to low: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Sodium, to low | 1 | 0
  7 Day Follow-up, Total bilirubin, to high: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Total bilirubin, to high | 1 | 0
  7 Day Follow-up, Total protein, to high: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Total protein, to high | 1 | 1
  7 Day Follow-up, Urea/BUN, to low: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Urea/BUN, to low | 1 | 1
  7 Day Follow-up, Urea/BUN, to high: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Urea/BUN, to high | 1 | 1
  7 Day Follow-up, Uric acid, to low: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Uric acid, to low | 1 | 1
  7 Day Follow-up, Uric acid, to high: number analyzed (Participants) | 45 | 24
  7 Day Follow-up, Uric acid, to high | 5 | 0
  28 Day Follow-up, ALT, to high: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, ALT, to high | 2 | 0
  28 Day Follow-up, ALP, to high: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, ALP, to high | 0 | 1
  28 Day Follow-up, AST, to high: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, AST, to high | 1 | 1
  28 Day Follow-up, Calcium, to low: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, Calcium, to low | 3 | 0
  28 Day Follow-up, Calcium, to high: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, Calcium, to high | 1 | 0
  28 Day Follow-up, CO2/bicarbonate, to low: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, CO2/bicarbonate, to low | 1 | 6
  28 Day Follow-up, Chloride, to low: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, Chloride, to low | 0 | 1
  28 Day Follow-up, Chloride, to high: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, Chloride, to high | 2 | 3
  28 Day Follow-up, Creatine kinase, to high: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, Creatine kinase, to high | 5 | 2
  28 Day Follow-up, Creatinine, to low: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, Creatinine, to low | 2 | 3
  28 Day Follow-up, Creatinine, to high: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, Creatinine, to high | 1 | 0
  28 Day Follow-up, GGT, to high: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, GGT, to high | 1 | 1
  28 Day Follow-up, Glucose, to high: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, Glucose, to high | 7 | 3
  28 Day Follow-up, Potassium, to low: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, Potassium, to low | 2 | 1
  28 Day Follow-up, Sodium, to low: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, Sodium, to low | 0 | 2
  28 Day Follow-up, Total protein, to low: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, Total protein, to low | 2 | 0
  28 Day Follow-up, Total protein, to high: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, Total protein, to high | 1 | 0
  28 Day Follow-up, Urea/BUN, to low: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, Urea/BUN, to low | 1 | 0
  28 Day Follow-up, Uric acid, to low: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, Uric acid, to low | 0 | 2
  28 Day Follow-up, Uric acid, to high: number analyzed (Participants) | 40 | 23
  28 Day Follow-up, Uric acid, to high | 1 | 0

24. Primary Outcome: Number of Participants With Abnormal Transition From Baseline in Hematology Values Relative to Normal Range
Description: The parameters of clinical chemistry included basophils, eosinophils, lymphocytes, monocytes, total neutrophils, WBC count, platelet count, MCV, hemoglobin, MCHC, MCH, RBC count and reticulocyte count. The assessments were done at Day 1, Day 4, Day 8, Day 11, 7 Day Follow-up and 28 Day Follow-up. Baseline was defined as the assessment done on Day 1 (pre-dose). Data is reported for number of participants with abnormal transition from Baseline 'to high' or 'to low' relative to normal range. Only those parameters for which at least one value of abnormal transition was reported are summarized.
Time Frame: Day 1 (pre-dose, Baseline) up Follow-up (28 Day Follow-up, Day 40)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Participants
  Day 4, Eosinophils, to low: number analyzed (Participants) | 44 | 25
  Day 4, Eosinophils, to low | 6 | 1
  Day 4, Eosinophils, to high: number analyzed (Participants) | 44 | 25
  Day 4, Eosinophils, to high | 1 | 0
  Day 4, Hemoglobin, to low: number analyzed (Participants) | 44 | 25
  Day 4, Hemoglobin, to low | 3 | 3
  Day 4, Lymphocytes, to low: number analyzed (Participants) | 44 | 25
  Day 4, Lymphocytes, to low | 1 | 0
  Day 4, MCHC, to low: number analyzed (Participants) | 44 | 25
  Day 4, MCHC, to low | 2 | 0
  Day 4, Monocytes, to low: number analyzed (Participants) | 44 | 25
  Day 4, Monocytes, to low | 3 | 1
  Day 4, Monocytes, to high: number analyzed (Participants) | 44 | 25
  Day 4, Monocytes, to high | 0 | 1
  Day 4, Platelet count, to high: number analyzed (Participants) | 42 | 25
  Day 4, Platelet count, to high | 2 | 1
  Day 4, RBC count, to low: number analyzed (Participants) | 44 | 25
  Day 4, RBC count, to low | 2 | 4
  Day 4, Reticulocytes, to low: number analyzed (Participants) | 44 | 25
  Day 4, Reticulocytes, to low | 1 | 1
  Day 4, Reticulocytes, to high: number analyzed (Participants) | 44 | 25
  Day 4, Reticulocytes, to high | 2 | 1
  Day 4, Total neutrophils, to low: number analyzed (Participants) | 44 | 25
  Day 4, Total neutrophils, to low | 1 | 0
  Day 4, Total neutrophils, to high: number analyzed (Participants) | 44 | 25
  Day 4, Total neutrophils, to high | 1 | 0
  Day 4, WBC count, to low: number analyzed (Participants) | 44 | 25
  Day 4, WBC count, to low | 2 | 1
  Day 4, WBC count, to high: number analyzed (Participants) | 44 | 25
  Day 4, WBC count, to high | 1 | 0
  Day 8, Eosinophils, to low: number analyzed (Participants) | 44 | 24
  Day 8, Eosinophils, to low | 3 | 2
  Day 8, Hemoglobin, to low: number analyzed (Participants) | 44 | 24
  Day 8, Hemoglobin, to low | 1 | 2
  Day 8, Lymphocytes, to low: number analyzed (Participants) | 44 | 24
  Day 8, Lymphocytes, to low | 1 | 0
  Day 8, MCHC, to low: number analyzed (Participants) | 44 | 24
  Day 8, MCHC, to low | 1 | 0
  Day 8, MCV, to high: number analyzed (Participants) | 44 | 24
  Day 8, MCV, to high | 1 | 0
  Day 8, Monocytes, to low: number analyzed (Participants) | 44 | 24
  Day 8, Monocytes, to low | 3 | 0
  Day 8, Platelet count, to high: number analyzed (Participants) | 44 | 24
  Day 8, Platelet count, to high | 2 | 0
  Day 8, RBC count, to low: number analyzed (Participants) | 44 | 24
  Day 8, RBC count, to low | 1 | 2
  Day 8, Reticulocytes, to low: number analyzed (Participants) | 44 | 24
  Day 8, Reticulocytes, to low | 0 | 4
  Day 8, Reticulocytes, to high: number analyzed (Participants) | 44 | 24
  Day 8, Reticulocytes, to high | 5 | 2
  Day 8, Total neutrophils, to low: number analyzed (Participants) | 44 | 24
  Day 8, Total neutrophils, to low | 3 | 0
  Day 8, Total neutrophils, to high: number analyzed (Participants) | 44 | 24
  Day 8, Total neutrophils, to high | 0 | 1
  Day 8, WBC count, to low: number analyzed (Participants) | 44 | 24
  Day 8, WBC count, to low | 2 | 0
  Day 11, Eosinophils, to low: number analyzed (Participants) | 40 | 23
  Day 11, Eosinophils, to low | 2 | 1
  Day 11, Hemoglobin, to low: number analyzed (Participants) | 40 | 23
  Day 11, Hemoglobin, to low | 2 | 2
  Day 11, Hemoglobin, to high: number analyzed (Participants) | 40 | 23
  Day 11, Hemoglobin, to high | 1 | 0
  Day 11, Lymphocytes, to low: number analyzed (Participants) | 40 | 23
  Day 11, Lymphocytes, to low | 3 | 0
  Day 11, Monocytes, to low: number analyzed (Participants) | 40 | 23
  Day 11, Monocytes, to low | 5 | 1
  Day 11, Platelet count, to high: number analyzed (Participants) | 40 | 22
  Day 11, Platelet count, to high | 1 | 0
  Day 11, RBC count, to low: number analyzed (Participants) | 40 | 23
  Day 11, RBC count, to low | 2 | 1
  Day 11, Reticulocytes, to low: number analyzed (Participants) | 40 | 23
  Day 11, Reticulocytes, to low | 3 | 1
  Day 11, Reticulocytes, to high: number analyzed (Participants) | 40 | 23
  Day 11, Reticulocytes, to high | 3 | 4
  Day 11, Total neutrophils, to low: number analyzed (Participants) | 40 | 23
  Day 11, Total neutrophils, to low | 1 | 1
  Day 11, Total neutrophils, to high: number analyzed (Participants) | 40 | 23
  Day 11, Total neutrophils, to high | 1 | 0
  Day 11, WBC count, to low: number analyzed (Participants) | 40 | 23
  Day 11, WBC count, to low | 2 | 0
  Day 11, WBC count, to high: number analyzed (Participants) | 40 | 23
  Day 11, WBC count, to high | 1 | 0
  7 Day Follow-up, Eosinophils, to low: number analyzed (Participants) | 45 | 25
  7 Day Follow-up, Eosinophils, to low | 0 | 3
  7 Day Follow-up, Hemoglobin, to low: number analyzed (Participants) | 45 | 25
  7 Day Follow-up, Hemoglobin, to low | 1 | 1
  7 Day Follow-up, Lymphocytes, to low: number analyzed (Participants) | 45 | 25
  7 Day Follow-up, Lymphocytes, to low | 1 | 1
  7 Day Follow-up, Monocytes, to low: number analyzed (Participants) | 45 | 25
  7 Day Follow-up, Monocytes, to low | 5 | 1
  7 Day Follow-up, Platelet count, to low: number analyzed (Participants) | 45 | 25
  7 Day Follow-up, Platelet count, to low | 1 | 0
  7 Day Follow-up, RBC count, to low: number analyzed (Participants) | 45 | 25
  7 Day Follow-up, RBC count, to low | 2 | 1
  7 Day Follow-up, Reticulocytes, to low: number analyzed (Participants) | 45 | 25
  7 Day Follow-up, Reticulocytes, to low | 4 | 0
  7 Day Follow-up, Reticulocytes, to high: number analyzed (Participants) | 45 | 25
  7 Day Follow-up, Reticulocytes, to high | 1 | 10
  7 Day Follow-up, Total neutrophils, to low: number analyzed (Participants) | 45 | 25
  7 Day Follow-up, Total neutrophils, to low | 1 | 0
  7 Day Follow-up, Total neutrophils, to high: number analyzed (Participants) | 45 | 25
  7 Day Follow-up, Total neutrophils, to high | 1 | 1
  7 Day Follow-up, WBC count, to low: number analyzed (Participants) | 45 | 25
  7 Day Follow-up, WBC count, to low | 1 | 0
  7 Day Follow-up, WBC count, to high: number analyzed (Participants) | 45 | 25
  7 Day Follow-up, WBC count, to high | 1 | 1
  28 Day Follow-up, Eosinophils, to low: number analyzed (Participants) | 39 | 22
  28 Day Follow-up, Eosinophils, to low | 1 | 1
  28 Day Follow-up, Hemoglobin, to low: number analyzed (Participants) | 39 | 22
  28 Day Follow-up, Hemoglobin, to low | 1 | 3
  28 Day Follow-up, Hemoglobin, to high: number analyzed (Participants) | 39 | 22
  28 Day Follow-up, Hemoglobin, to high | 1 | 0
  28 Day Follow-up, Lymphocytes, to low: number analyzed (Participants) | 39 | 22
  28 Day Follow-up, Lymphocytes, to low | 1 | 0
  28 Day Follow-up, Lymphocytes, to high: number analyzed (Participants) | 39 | 22
  28 Day Follow-up, Lymphocytes, to high | 1 | 0
  28 Day Follow-up, MCHC, to low: number analyzed (Participants) | 39 | 22
  28 Day Follow-up, MCHC, to low | 1 | 0
  28 Day Follow-up, Monocytes, to low: number analyzed (Participants) | 39 | 22
  28 Day Follow-up, Monocytes, to low | 1 | 0
  28 Day Follow-up, Platelet count, to low: number analyzed (Participants) | 38 | 22
  28 Day Follow-up, Platelet count, to low | 0 | 1
  28 Day Follow-up, Platelet count, to high: number analyzed (Participants) | 38 | 22
  28 Day Follow-up, Platelet count, to high | 2 | 0
  28 Day Follow-up, RBC count, to low: number analyzed (Participants) | 39 | 22
  28 Day Follow-up, RBC count, to low | 0 | 4
  28 Day Follow-up, Reticulocytes, to low: number analyzed (Participants) | 39 | 22
  28 Day Follow-up, Reticulocytes, to low | 0 | 1
  28 Day Follow-up, Reticulocytes, to high: number analyzed (Participants) | 39 | 22
  28 Day Follow-up, Reticulocytes, to high | 3 | 4
  28 Day Follow-up, Total neutrophils, to low: number analyzed (Participants) | 39 | 22
  28 Day Follow-up, Total neutrophils, to low | 1 | 0
  28 Day Follow-up, Total neutrophils, to high: number analyzed (Participants) | 39 | 22
  28 Day Follow-up, Total neutrophils, to high | 1 | 1
  28 Day Follow-up, WBC count, to low: number analyzed (Participants) | 39 | 22
  28 Day Follow-up, WBC count, to low | 1 | 0
  28 Day Follow-up, WBC count, to high: number analyzed (Participants) | 39 | 22
  28 Day Follow-up, WBC count, to high | 2 | 1

25. Secondary Outcome: Number of Participants With Clinical Success of Clinical Response
Description: The clinical response was evaluated by the investigator at end of therapy (within 3 days post therapy; Day 12-14) and Follow-up (7 day Follow-up; Day 16 to 19 and 28 day Follow-up; Day 37 to 40). Clinical response was determined after clinical evaluation of reviewing clinical signs and symptoms. Clinical success was defined as total resolution of all signs and symptoms of infection recorded at Baseline, or improvement to such an extent that no further antimicrobial therapy was necessary, including a pus/exudate skin infection score (SIS) of 0.
Time Frame: Up to Follow-up (28 Day Follow-up, Day 40)
Population: Intent-to-Treat Clinical (ITTC) Population was defined as all randomized participants who received at least one dose of study medication. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Participants
  Day 11: number analyzed (Participants) | 41 | 24
  Day 11 | 38 | 24
  7 Day Follow-up: number analyzed (Participants) | 44 | 25
  7 Day Follow-up | 38 | 25
  28 Day Follow-up: number analyzed (Participants) | 41 | 23
  28 Day Follow-up | 37 | 23

26. Secondary Outcome: Percentage of Participants With Clinical Success of Clinical Outcome
Description: The clinical response was determined by the investigator after clinical evaluation of reviewing clinical signs and symptoms at end of therapy (within 3 days post therapy; visit window of Day 12-14) and 7 day Follow-up ( visit window of Day 16 to 19), and the resulting clinical outcome was assigned, for each participant. Clinical success was defined as total resolution of all signs and symptoms of infection recorded at Baseline, or improvement to such an extent that no further antimicrobial therapy was necessary, including a pus/exudates SIS of 0.
Time Frame: Day 11 (end of therapy) and Follow-up (7 Day Follow-up, Day 19)
Population: ITTC Population.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Percentage of participants
  End of therapy | 66.7 | 88.9
  Follow-up | 64.9 | 88.9
Statistical Analysis 1: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for end of therapy Clinical Success; Test type: Superiority or Other; Regression, Logistic; Difference = -22.2
Statistical Analysis 2: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Follow-up Clinical Success; Test type: Superiority or Other; Regression, Logistic; Difference = -24.0

27. Secondary Outcome: Percentage of Participants With Microbiological Success of Microbiological Outcome at End of Therapy
Description: The 'by pathogen' microbiological response was determined by comparing the Baseline (Day 1) culture results to the culture results at the end of therapy (visit window of Day 12-14), and the corresponding microbiological outcome (success or failure) by participant was then assigned. Microbiological success was defined as: elimination of Baseline pathogens (defined as microbiological eradication in microbiological response); clinical outcome was success such that no culture was obtained due to lack of culturable material, secondary to adequate clinical response, and was documented in the electronic case report form (eCRF) (defined as presumed microbiological eradication in microbiological response); new pathogen not previously identified, was identified at end of therapy in a participant who was a 'clinical success' (defined as colonization in microbiological response).
Time Frame: Day 11 (end of therapy)
Population: Intent-to-Treat Bacteriology (ITTB) Population was defined as all randomized participants who received at least one dose of study medication and who had a pathogen isolated at Baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 37 | 18
Percentage of participants | 59.5 | 94.4
Statistical Analysis 1: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; Test type: Superiority or Other; Regression, Logistic; Difference = -35.0, 95% CI 2-sided [-60.6 to -9.4]

28. Secondary Outcome: Percentage of Participants With Microbiological Success of Microbiological Outcome at Follow-up
Description: The 'by pathogen' microbiological response was determined by comparing the Baseline (Day 1) culture results to culture results at Follow-up (Day 16-19), and corresponding microbiological outcome (success or failure) by participant was then assigned. Microbiological success was defined as: Baseline pathogen was eradicated or presumed eradicated at end of therapy, or Baseline pathogens were present at end of therapy and is absent at Follow-up (microbiological eradication in microbiological response); Baseline pathogen was eradicated or presumed eradicated at end of therapy, or the Baseline pathogens were present at end of therapy and, participant was a 'clinical success', such that no culture was obtained due to lack of culturable material, secondary to adequate clinical response, and was documented in the eCRF (microbiological eradication); a new pathogen, not previously identified at Baseline, was identified at Follow-up in a participant who was a 'clinical success' (colonization)
Time Frame: Follow-up (7 Day Follow-up, Day 19)
Population: ITTB Population.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 37 | 18
Percentage of participants | 59.5 | 94.4
Statistical Analysis 1: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; Test type: Superiority or Other; Regression, Logistic; Difference = -35.0, 95% CI 2-sided [-60.6 to -9.4]

29. Secondary Outcome: Percentage of Participants With Therapeutic Success of Therapeutic Outcome
Description: Therapeutic outcome was combined clinical and microbiological outcome. Therapeutic outcome was a measure of the overall efficacy response, and a therapeutic success referred to participants who had been deemed both a 'clinical success' and a 'microbiological success'. All other combinations (other than 'clinical success' + 'microbiological success') were deemed failures for therapeutic outcome. Therapeutic outcome was determined programmatically, obtained at 7 day Follow-up.
Time Frame: Follow-up (7 day Follow-up, Day 19)
Population: Per Protocol Bacteriology (PPB) Population was defined as ITTB participants who adhered to protocol-specific criteria (i.e., no protocol violation ): taking 80% of medications and/or not missing more than 48 h in a row of study drug, and have both end of therapy and 7 day Follow-up to be evaluable and a documented pathogen cultured at Baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 22 | 17
Percentage of participants | 0.8636 [0.7202 to 1.0000] | 1.0000 [1.0000 to 1.0000]

30. Secondary Outcome: Mean Short Form McGill Pain Questionnaire-2 (SF-MPQ-2) Sub-score of Continuous Pain, Intermittent Pain, Neuropathic Pain and Affective Descriptors at Indicated Time Points
Description: SF-MPQ-2 is composed of 22 items that describes different quantities of pain and related symptoms. Sub-score of continuous pain represents mean of throbbing pain, cramping pain, gnawing pain, aching pain, heavy pain and tender (mean of items 1, 5, 6, 8, 9 and 10). Sub-score of intermittent pain represents mean of shooting pain, stabbing pain, sharp pain, splitting pain, electric-shock pain and piercing (mean of items 2, 3, 4, 11, 16 and 18). Sub-score of neuropathic pain represents mean of hot-burning pain, cold-freezing pain, pain caused by light touch, itching, tingling or pins and needles, numbness (mean of items 7, 17, 19, 20, 21 and 22). Sub-score of affective descriptors represents mean of tiring-exhaustive, sickening, fearful, punishing-cruel (mean of items 12, 13, 14 and 15). Scores ranged from 0 to 10, where 0 indicated absence of symptom and higher score indicated more severe symptoms. Assessments were done at Day 1, Day 2, Day 3, Day 4, Day 8, Day 11 and 7 Day Follow-up.
Time Frame: Up to Follow-up (7 Day Follow up, Day 19)
Population: ITTC Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Scores on scale
  Continuous Pain, Day 1 | 4.459 (2.8567) | 4.889 (2.2773)
  Continuous Pain, Day 2: number analyzed (Participants) | 52 | 25
  Continuous Pain, Day 2 | 3.407 (2.4454) | 3.533 (2.6745)
  Continuous Pain, Day 3: number analyzed (Participants) | 48 | 26
  Continuous Pain, Day 3 | 2.826 (2.5509) | 2.744 (2.8477)
  Continuous Pain, Day 4: number analyzed (Participants) | 46 | 25
  Continuous Pain, Day 4 | 2.645 (2.7701) | 2.067 (2.4462)
  Continuous Pain, Day 8: number analyzed (Participants) | 44 | 24
  Continuous Pain, Day 8 | 1.420 (1.9653) | 1.389 (2.0534)
  Continuous Pain, Day 11: number analyzed (Participants) | 41 | 24
  Continuous Pain, Day 11 | 0.882 (1.3387) | 0.806 (1.3976)
  Continuous Pain, 7 Day Follow-up: number analyzed (Participants) | 43 | 25
  Continuous Pain, 7 Day Follow-up | 0.733 (1.3018) | 0.533 (1.2342)
  Intermittent Pain, Day 1 | 3.836 (3.1349) | 3.802 (2.9067)
  Intermittent Pain, Day 2: number analyzed (Participants) | 52 | 25
  Intermittent Pain, Day 2 | 2.337 (2.4214) | 2.693 (2.9867)
  Intermittent Pain, Day 3: number analyzed (Participants) | 49 | 26
  Intermittent Pain, Day 3 | 2.078 (2.4989) | 2.244 (2.7913)
  Intermittent Pain, Day 4: number analyzed (Participants) | 46 | 25
  Intermittent Pain, Day 4 | 1.906 (2.6239) | 1.620 (2.4188)
  Intermittent Pain, Day 8: number analyzed (Participants) | 44 | 24
  Intermittent Pain, Day 8 | 0.871 (1.8040) | 1.236 (1.9640)
  Intermittent Pain, Day 11: number analyzed (Participants) | 41 | 24
  Intermittent Pain, Day 11 | 0.504 (0.9927) | 0.688 (1.4902)
  Intermittent Pain, 7 Day Follow-up: number analyzed (Participants) | 43 | 25
  Intermittent Pain, 7 Day Follow-up | 0.581 (1.3429) | 0.440 (1.1656)
  Neuropathic Pain, Day 1 | 3.520 (2.5554) | 3.846 (2.3705)
  Neuropathic Pain, Day 2: number analyzed (Participants) | 52 | 25
  Neuropathic Pain, Day 2 | 2.705 (2.0982) | 2.193 (2.2632)
  Neuropathic Pain, Day 3: number analyzed (Participants) | 49 | 26
  Neuropathic Pain, Day 3 | 2.327 (2.0089) | 2.026 (2.3526)
  Neuropathic Pain, Day 4: number analyzed (Participants) | 46 | 25
  Neuropathic Pain, Day 4 | 2.391 (2.3476) | 1.613 (2.0473)
  Neuropathic Pain, Day 8: number analyzed (Participants) | 44 | 24
  Neuropathic Pain, Day 8 | 1.508 (1.7878) | 1.410 (2.0042)
  Neuropathic Pain, Day 11: number analyzed (Participants) | 41 | 24
  Neuropathic Pain, Day 11 | 0.813 (1.1113) | 0.778 (1.2450)
  Neuropathic Pain, 7 Day Follow-up: number analyzed (Participants) | 42 | 25
  Neuropathic Pain, 7 Day Follow-up | 0.690 (1.1515) | 0.593 (1.1707)
  Affective Descriptors, Day 1 | 3.360 (3.0063) | 2.806 (2.9000)
  Affective Descriptors, Day 2: number analyzed (Participants) | 52 | 25
  Affective Descriptors, Day 2 | 2.226 (2.5925) | 2.500 (2.9244)
  Affective Descriptors, Day 3: number analyzed (Participants) | 49 | 26
  Affective Descriptors, Day 3 | 1.929 (2.4088) | 1.692 (2.6517)
  Affective Descriptors, Day 4: number analyzed (Participants) | 46 | 25
  Affective Descriptors, Day 4 | 1.641 (2.4736) | 1.330 (2.2287)
  Affective Descriptors, Day 8: number analyzed (Participants) | 44 | 24
  Affective Descriptors, Day 8 | 0.852 (1.5970) | 1.021 (2.0811)
  Affective Descriptors, Day 11: number analyzed (Participants) | 41 | 24
  Affective Descriptors, Day 11 | 0.640 (1.1320) | 0.490 (1.2079)
  Affective Descriptors, 7 Day Follow-up: number analyzed (Participants) | 43 | 25
  Affective Descriptors, 7 Day Follow-up | 0.483 (1.0400) | 0.430 (1.1099)

31. Secondary Outcome: Mean Exudate or Pus Sub-score of SIS at Indicated Time Points
Description: The SIS consist of 7 items of exudate or pus, crusting, erythema or inflammation, tissue warmth, tissue edema, itching and pain. The exudate or pus sub-score of SIS was rated on a 7-point scale ranging from 0 to 6, where 0 indicated absence of symptom and 6 indicated severe symptom. Assessments were done at Day 1, Day 2, Day 3, Day 4, Day 8, Day 11, 7 Day Follow-up and 28 Day Follow-up.
Time Frame: Up to Follow-up (28 Day Follow-up, Day 40)
Population: ITTC Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Scores on scale
  Day 1 | 3.2 (2.23) | 3.2 (2.39)
  Day 2: number analyzed (Participants) | 51 | 25
  Day 2 | 3.0 (1.81) | 2.8 (1.97)
  Day 3: number analyzed (Participants) | 49 | 26
  Day 3 | 2.1 (1.56) | 2.2 (1.86)
  Day 4: number analyzed (Participants) | 46 | 25
  Day 4 | 1.5 (1.60) | 1.7 (1.51)
  Day 8: number analyzed (Participants) | 44 | 24
  Day 8 | 0.8 (1.29) | 0.4 (0.71)
  Day 11: number analyzed (Participants) | 41 | 24
  Day 11 | 0.2 (0.70) | 0.0 (0.00)
  7 Day Follow-up: number analyzed (Participants) | 43 | 25
  7 Day Follow-up | 0.1 (0.37) | 0.0 (0.00)
  28 Day Follow-up: number analyzed (Participants) | 41 | 23
  28 Day Follow-up | 0.0 (0.00) | 0.0 (0.00)
Statistical Analysis 1: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 2 exudate or pus score; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.41 to 0.74]
Statistical Analysis 2: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 3 exudate or pus score; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.70 to 0.45] — The point estimate was calculated as least square mean difference (final values) of GSK1322322 1500 mg and Linezolid 600 mg
Statistical Analysis 3: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 4 exudate or pus score; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.74 to 0.43] — [estimate comment as in outcome 31, analysis 2]
Statistical Analysis 4: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 8 exudate or pus score; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-0.25 to 0.95] — [estimate comment as in outcome 31, analysis 2]
Statistical Analysis 5: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 11 exudate or pus score; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.49 to 0.72] — [estimate comment as in outcome 31, analysis 2]
Statistical Analysis 6: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for 7 Day Follow- up exudate or pus score; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.53 to 0.66] — [estimate comment as in outcome 31, analysis 2]
Statistical Analysis 7: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for 28 Day Follow- up exudate or pus score; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.65 to 0.58] — [estimate comment as in outcome 31, analysis 2]

32. Secondary Outcome: Mean Total SIS at Indicated Time Points
Description: The investigator evaluated the infection by grading the infected lesion according to SIS. The SIS consist of 7 items of exudate or pus, crusting, erythema or inflammation, tissue warmth, tissue edema, itching and pain. The items were rated on a 7-point scale ranging from 0 to 6, where 0 indicated absence of symptom and 6 indicated severe symptom. The total score ranged from 0 to 42, where 0 indicated absence of symptoms and higher score indicated more severe symptoms. Assessments were done at Day 1, Day 2, Day 3, Day 4, Day 8, Day 11, 7 Day Follow-up and 28 Day Follow-up.
Time Frame: Up to Follow-up (28 Day Follow-up, Day 40)
Population: ITTC Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Scores on scale
  Day 1 | 25.7 (5.44) | 26.0 (4.39)
  Day 2: number analyzed (Participants) | 51 | 25
  Day 2 | 22.2 (5.24) | 23.3 (5.01)
  Day 3: number analyzed (Participants) | 49 | 26
  Day 3 | 17.2 (6.09) | 18.1 (6.59)
  Day 4: number analyzed (Participants) | 46 | 25
  Day 4 | 14.6 (6.47) | 14.1 (6.19)
  Day 8: number analyzed (Participants) | 44 | 24
  Day 8 | 8.8 (5.52) | 6.9 (4.17)
  Day 11: number analyzed (Participants) | 41 | 24
  Day 11 | 3.7 (3.53) | 2.3 (2.11)
  7 Day Follow-up: number analyzed (Participants) | 43 | 25
  7 Day Follow-up | 2.4 (2.55) | 1.8 (2.07)
  28 Day Follow-up: number analyzed (Participants) | 41 | 23
  28 Day Follow-up | 0.3 (1.29) | 0.1 (0.34)
Statistical Analysis 1: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 2 total SIS; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Net) = -0.86, 95% CI 2-sided [-3.04 to 1.33] — [estimate comment as in outcome 31, analysis 2]
Statistical Analysis 2: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 3 total SIS; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-2.94 to 1.41] — [estimate comment as in outcome 31, analysis 2]
Statistical Analysis 3: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 4 total SIS; Test type: Superiority or Other; Mean Difference (Final Values) = 0.54, 95% CI 2-sided [-1.68 to 2.75] — [estimate comment as in outcome 31, analysis 2]
Statistical Analysis 4: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 8 total SIS; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.79, 95% CI 2-sided [-0.46 to 4.05] — [estimate comment as in outcome 31, analysis 2]
Statistical Analysis 5: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 11 total SIS; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.19, 95% CI 2-sided [-1.09 to 3.47] — [estimate comment as in outcome 31, analysis 2]
Statistical Analysis 6: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for 7 Day Follow-up total SIS; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [-1.49 to 2.98] — [estimate comment as in outcome 31, analysis 2]
Statistical Analysis 7: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for 28 Day Follow-up total SIS; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-2.09 to 2.52] — [estimate comment as in outcome 31, analysis 2]

33. Secondary Outcome: Mean Change From Baseline in Total SIS at Indicated Time Points
Description: The investigator evaluated the infection by grading the infected lesion according to SIS. The SIS consist of 7 items of exudate or pus, crusting, erythema or inflammation, tissue warmth, tissue edema, itching and pain. The items were rated on a 7-point scale ranging from 0 to 6, where 0 indicated absence of symptom and 6 indicated severe symptom. The total score ranged from 0 to 42, where 0 indicated absence of symptoms and higher score indicated more severe symptoms. Baseline was defined as the assessment value done on Day 1. The change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 1, Day 2, Day 3, Day 4, Day 8, Day 11, 7 Day Follow-up and 28 Day Follow-up) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to missing as well.
Time Frame: Day 1 (Baseline ) up to Follow-up (28 Day Follow-up, Day 40)
Population: ITTC Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Scores on scale
  Day 2: number analyzed (Participants) | 51 | 25
  Day 2 | -3.4 (4.83) | -3.1 (4.98)
  Day 3: number analyzed (Participants) | 49 | 26
  Day 3 | -8.4 (6.39) | -8.0 (6.79)
  Day 4: number analyzed (Participants) | 46 | 25
  Day 4 | -10.9 (6.98) | -11.9 (6.84)
  Day 8: number analyzed (Participants) | 44 | 24
  Day 8 | -16.8 (7.22) | -19.0 (6.38)
  Day 11: number analyzed (Participants) | 41 | 24
  Day 11 | -22.0 (6.06) | -23.6 (4.82)
  7 Day Follow-up: number analyzed (Participants) | 43 | 25
  7 Day Follow-up | -23.0 (5.91) | -24.2 (4.75)
  28 Day Follow-up: number analyzed (Participants) | 41 | 23
  28 Day Follow-up | -25.1 (5.54) | -26.1 (3.98)
Statistical Analysis 1: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 2 total SIS; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Net) = -0.86, 95% CI 2-sided [-3.04 to 1.33] — The point estimate was calculated as least square mean difference (net values) of GSK1322322 1500 mg and Linezolid 600 mg
Statistical Analysis 2: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 3 total SIS; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Net) = -0.77, 95% CI 2-sided [-2.94 to 1.41] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 3: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 4 total SIS; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Net) = 0.54, 95% CI 2-sided [-1.68 to 2.75] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 4: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 8 total SIS; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Net) = 1.79, 95% CI 2-sided [-0.46 to 4.05] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 5: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 11 total SIS; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Net) = 1.19, 95% CI 2-sided [-1.09 to 3.47] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 6: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for 7 Day Follow-up total SIS; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Net) = 0.74, 95% CI 2-sided [-1.49 to 2.98] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 7: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for 28 Day Follow-up total SIS; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Net) = 0.21, 95% CI 2-sided [-2.09 to 2.52] — [estimate comment as in outcome 33, analysis 1]

34. Secondary Outcome: Mean Change From Baseline in Wound Area at Indicated Time Points
Description: The area of the infected lesion size was calculated as the product between the length (L) and width (W) of the lesion size. The wound was measured by the investigator in centimeters (cm), using a standard metric ruler. Baseline was defined as the assessment value done on Day 1. The change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 1, Day 2, Day 3, Day 4, Day 8, Day 11, 7 Day Follow-up and 28 Day Follow-up) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to missing as well.
Time Frame: Day 1 (Baseline) up to Follow-up (28 Day Follow-up, Day 40)
Population: ITTC Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
cm^2
  Day 2: number analyzed (Participants) | 51 | 25
  Day 2 | -23.22 (52.486) | -20.71 (88.184)
  Day 3: number analyzed (Participants) | 49 | 26
  Day 3 | -67.69 (93.511) | -124.27 (188.568)
  Day 4: number analyzed (Participants) | 46 | 25
  Day 4 | -119.96 (86.544) | -209.79 (224.125)
  Day 8: number analyzed (Participants) | 44 | 24
  Day 8 | -192.92 (175.606) | -291.86 (338.675)
  Day 11: number analyzed (Participants) | 41 | 24
  Day 11 | -234.99 (276.801) | -329.93 (362.831)
  7 Day Follow-up: number analyzed (Participants) | 43 | 25
  7 Day Follow-up | -231.32 (273.285) | -335.20 (363.233)
  28 Day Follow-up: number analyzed (Participants) | 41 | 23
  28 Day Follow-up | -242.92 (277.312) | -344.99 (383.444)
Statistical Analysis 1: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 2 wound area; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Net) = -68.85, 95% CI 2-sided [-132.8 to -4.95] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 2: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 3 wound area; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Net) = -3.06, 95% CI 2-sided [-66.54 to 60.43] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 3: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 4 wound area; Test type: Superiority or Other; Mixed Models Analysis; Median Difference (Net) = 31.47, 95% CI 2-sided [-33.53 to 96.47] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 4: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 8 wound area; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Net) = 43.94, 95% CI 2-sided [-22.43 to 110.31] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 5: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Day 11 wound area; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Net) = 34.21, 95% CI 2-sided [-33.03 to 101.45] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 6: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for 7 Day Follow-up wound area; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Net) = 37.57, 95% CI 2-sided [-28.25 to 103.40] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 7: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for 28 Day Follow-up wound area; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Net) = 37.40, 95% CI 2-sided [-30.77 to 105.56] — [estimate comment as in outcome 33, analysis 1]

35. Secondary Outcome: Percentage of Participants With Clinical Success at End of Therapy by Pathogen Isolated at Baseline
Description: Clinical success was defined as total resolution of all signs and symptoms of infection recorded at Baseline, or improvement to such an extent that no further antimicrobial therapy was necessary, including a pus/exudates SIS of 0. The pathogens isolated at Baseline included staphylococcus aureus (methicillin-resistant staphylococcus aureus [MRSA] and methicillin-susceptible staphylococcus aureus [MSSA] as defined by susceptibility to cefoxitin or oxacilin), streptococcus pyogenes, other streptococcus species, other Gram-positive pathogens and Gram-negative pathogens. Data is categorized for the percentage of participants with clinical success for each of the pathogens, all pathogens and no pathogens.
Time Frame: Up to Follow-up (28 Day Follow-up, Day 40)
Population: ITTC Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
Number analyzed (Participants) | 57 | 27
Percentage of participants
  Staphylococcus aureus (all): number analyzed (Participants) | 36 | 16
  Staphylococcus aureus (all) | 58.3 | 93.8
  MRSA: number analyzed (Participants) | 22 | 8
  MRSA | 50.0 | 87.5
  MSSA: number analyzed (Participants) | 14 | 8
  MSSA | 71.4 | 100.0
  Streptococcus pyogenes: number analyzed (Participants) | 3 | 1
  Streptococcus pyogenes | 33.3 | 100.0
  Other Streptococcus species: number analyzed (Participants) | 0 | 1
  Other Streptococcus species |  | 100.0
  Other Gram-positive pathogens: number analyzed (Participants) | 0 | 1
  Other Gram-positive pathogens |  | 100.0
  Gram-negative pathogens: number analyzed (Participants) | 4 | 4
  Gram-negative pathogens | 75.0 | 100.0
  All pathogens: number analyzed (Participants) | 43 | 23
  All pathogens | 58.1 | 95.7
  No pathogens: number analyzed (Participants) | 20 | 9
  No pathogens | 80.0 | 77.8
Statistical Analysis 1: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Staphylococcus aureus (all); Test type: Superiority or Other; Regression, Logistic; Difference = -35.4
Statistical Analysis 2: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for MRSA; Test type: Superiority or Other; Regression, Logistic; Difference = -37.5
Statistical Analysis 3: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for MSSA; Test type: Superiority or Other; Regression, Logistic; Difference = -28.6
Statistical Analysis 4: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Streptococcus pyogenes; Test type: Superiority or Other; Regression, Logistic; Difference = -66.7
Statistical Analysis 5: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for Gram-negative pathogens; Test type: Superiority or Other; Regression, Logistic; Difference = -25.0
Statistical Analysis 6: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for All pathogens; Test type: Superiority or Other; Regression, Logistic; Difference = -37.5
Statistical Analysis 7: Comparison: GSK1322322 1500 mg BID vs Linezolid 600 mg BID; GSK1322322 1500 mg versus Linezolid 600 mg for No pathogens; Test type: Superiority or Other; Regression, Logistic; Difference = 2.2

36. Secondary Outcome: Population Pharmacokinetic Parameters of Apparent Total Clearance of GSK1322322 From Plasma After Oral Administration (CL/F)
Description: Blood samples were planned to be collected on Day 1, 0.25-1.5 hours post-initial dose (corresponding to the safety laboratory and ECG timepoint), and 1.5-3 hours post-initial dose (corresponding to the safety laboratory and ECG timepoint), and Day 4, 4-12 hours post-morning dose (corresponding to the safety laboratory and ECG timepoint), and Day 8, pre-morning dose (corresponding to safety laboratory and ECG timepoint) during the outpatient visit. The data for this outcome measure was not collected and assessed.
Time Frame: Day 1 (0.25-1.5 hours post-initial dose, 1.5-3 hours post-initial dose), Day 4 (4-12 hours post-morning dose) and Day 8 (pre-morning dose)
Population: Pharmacokinetic (PK) Concentration Population defined all Participants in the "Safety Population" who underwent plasma PK sampling during the study and from whom a measurable plasma concentration above the assay's limit of quantification were obtained for one of the treatment regimens. No participants were analyzed for this outcome measure.
Arm/Group | GSK1322322 1500 mg BID
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs were collected up to Follow-up (28 Day Follow-up, Day 40)
Description: Safety Population was used.
Arm/Group | GSK1322322 1500 mg BID | Linezolid 600 mg BID
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/57 | 1/27
Other Adverse Events (participants affected / at risk) | 38/57 | 16/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1322322 1500 mg BID (N=57) | Linezolid 600 mg BID (N=27)
Multiple drug overdose (Injury, poisoning and procedural complications) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1322322 1500 mg BID (N=57) | Linezolid 600 mg BID (N=27)
Nausea (Gastrointestinal disorders) | 14 | 4
Diarrhoea (Gastrointestinal disorders) | 8 | 2
Vomiting (Gastrointestinal disorders) | 9 | 1
Flatulence (Gastrointestinal disorders) | 0 | 2
Blood glucose increased (Investigations) | 6 | 3
Alanine aminotransferase increased (Investigations) | 4 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 2
Haemoglobin decreased (Investigations) | 3 | 0
Headache (Nervous system disorders) | 7 | 2
Dizziness (Nervous system disorders) | 5 | 1
Fatigue (General disorders) | 3 | 0
Pain (General disorders) | 3 | 0
Pyrexia (General disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0
Skin infection (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.